CLINICAL TRIAL: NCT04147715
Title: A Phase 1, Randomized, Double-Blind, Single-Ascending-Dose, and Food Effect Study to Assess the Safety, Tolerability, Ventricular Repolarization, and Pharmacokinetics of S-648414 in Healthy Adult Study Participants (Part 1); A Phase 1, Randomized, Double-Blind, Multiple-Ascending-Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of S-648414 and A Drug-Drug Interaction Study With the CYP3A Substrate, Midazolam, in Healthy Adult Study Participants (Part 2)
Brief Title: Evaluation of Safety, Tolerability, Pharmacokinetics, Drug-Drug and Food Interactions of Single and Multiple Doses of S-648414 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 1908T0911
Record Dates: First submitted 2019-10-28; First posted 2019-11-01 (Actual); Results first posted 2021-10-20 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Healthy Volunteer
Keywords: Pharmacokinetics; S-648414; Food effect; Antiretroviral; Drug-drug interaction
MeSH Terms: interventions — Midazolam; dolutegravir

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Parts 1 and 2 were blinded studies. Part 3 was an open-label study and, therefore, did not include blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Part 1: Placebo (Placebo Comparator): Participants received a single oral dose of matching placebo in a fasted state on Day 1.
  Interventions: Drug: Placebo
- Part 1: 10 mg S-648414 (Experimental): Participants received a single oral dose of 10 mg S-648414 in a fasted state on Day 1.
  Interventions: Drug: S-648414
- Part 1: 30 mg S-648414 (Experimental): Participants received a single oral dose of 30 mg S-648414 in a fasted state on Day 1.
  Interventions: Drug: S-648414
- Part 1: 100 mg S-648414 (Experimental): Participants received a single oral dose of 100 mg S-648414 in a fasted state on Day 1 followed by a single dose of S-648414 in a fed state (after a high-fat meal) on Day 14.
  Interventions: Drug: S-648414
- Part 1: 250 mg S-648414 (Experimental): Participants received a single oral dose of 250 mg S-648414 in a fasted state on Day 1.
  Interventions: Drug: S-648414
- Part 1: 500 mg S-648414 (Experimental): Participants received a single oral dose of 500 mg S-648414 in a fasted state on Day 1.
  Interventions: Drug: S-648414
- Part 1: 1000 mg S-648414 (Experimental): Participants received a single oral dose of 1000 mg S-648414 in a fasted state on Day 1.
  Interventions: Drug: S-648414
- Part 2: Placebo + Midazolam (Placebo Comparator): Participants received matching placebo once a day on Days 1 to 14 and a single oral dose of 5 mg midazolam alone on Day -2 and co-administered with the placebo dose on Day 14.
  Interventions: Drug: Placebo; Drug: Midazolam
- Part 2: 50 mg S-648414 + Midazolam (Experimental): Participants received 50 mg S-648414 once a day on Days 1 to 14 and a single oral dose of 5 mg midazolam alone on Day -2 and co-administered with the S-648414 dose on Day 14.
  Interventions: Drug: S-648414; Drug: Midazolam
- Part 2: 30 mg S-648414 + Midazolam (Experimental): Participants received 30 mg S-648414 once a day on Days 1 to 14 and a single oral dose of 5 mg midazolam alone on Day -2 and co-administered with the S-648414 dose on Day 14.
  Interventions: Drug: S-648414; Drug: Midazolam
- Part 3: 100 mg S-648414 + Dolutegravir (Experimental): Participants received 50 mg dolutegravir orally once a day on Days 1 to 7, 100 mg S-648414 orally once a day on Days 15 to 21, and 50 mg dolutegravir co-administered with 100 mg S-648414 orally once a day on Days 22 to 28.
  Interventions: Drug: S-648414; Drug: Dolutegravir
- Part 3: 200 mg S-648414 + Dolutegravir (Experimental): Participants received 50 mg dolutegravir orally once a day on Days 1 to 7, 200 mg S-648414 orally once a day on Days 15 to 21, and 50 mg dolutegravir co-administered with 200 mg S-648414 orally once a day on Days 22 to 28.
  Interventions: Drug: S-648414; Drug: Dolutegravir

INTERVENTIONS:
Drug: S-648414 — Tablet for oral administration
  Arms: Part 1: 10 mg S-648414; Part 1: 100 mg S-648414; Part 1: 1000 mg S-648414; Part 1: 250 mg S-648414; Part 1: 30 mg S-648414; Part 1: 500 mg S-648414; Part 2: 30 mg S-648414 + Midazolam; Part 2: 50 mg S-648414 + Midazolam; Part 3: 100 mg S-648414 + Dolutegravir; Part 3: 200 mg S-648414 + Dolutegravir
Drug: Placebo — Tablet for oral administration
  Arms: Part 1: Placebo; Part 2: Placebo + Midazolam
Drug: Midazolam — Solution for oral administration
  Other Names: Versed
  Arms: Part 2: 30 mg S-648414 + Midazolam; Part 2: 50 mg S-648414 + Midazolam; Part 2: Placebo + Midazolam
Drug: Dolutegravir — Tablet for oral administration
  Other Names: TIVICAY
  Arms: Part 3: 100 mg S-648414 + Dolutegravir; Part 3: 200 mg S-648414 + Dolutegravir

SUMMARY:
The primary objective of Part 1 of the study is to evaluate the safety and tolerability of S-648414 after administration of a single oral dose of S-648414 in healthy adult study participants.

The primary objective of Part 2 is to evaluate the safety and tolerability of S-648414 after administration of multiple oral doses of S-648414 in healthy adult study participants.

The primary objectives of Part 3 are evaluate the safety and tolerability of S-648414 after administration of multiple oral doses of S-648414 in healthy adult study participants, and to evaluate the effect of S-648414 on the pharmacokinetics (PK) of dolutegravir and the effect of dolutegravir on the PK of S-648414 in healthy adult study participants.

DETAILED DESCRIPTION:
Amendment 2 of the study Protocol added a third part (Part 3) to the study. The revised Official Title for the Protocol is:

"A Phase 1, Randomized, Double-Blind, Single-Ascending-Dose, and Food Effect Study to Assess the Safety, Tolerability, Ventricular Repolarization, and Pharmacokinetics of S-648414 in Healthy Adult Study Participants (Part 1); A Phase 1, Randomized, Double-Blind, Multiple-Ascending-Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of S-648414 and A Drug-Drug Interaction Study with the CYP3A Substrate, Midazolam, in Healthy Adult Study Participants (Part 2); and A Phase 1 Open-Label Study to Assess the Effect of S-648414 on the Pharmacokinetics of Dolutegravir and the Effect of Dolutegravir on the Pharmacokinetics of S-648414 in Healthy Adult Study Participants (Part 3)"

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults ≥ 18 years in USA or ≥ 20 years in Japan to ≤ 55 years of age, at the time of signing the informed consent form (ICF).

   a) Specific to Japan sites: enrollment in Part 3 (Group I and J) will consist of only White or Black or African American race.
2. Capable of giving signed informed consent
3. Body mass index (BMI) ≥ 18.5 to < 32.0 kg/m² at the Screening visit．
4. Considered medically healthy as determined by the investigator or subinvestigator (suitably qualified), based on medical history and clinical evaluations including physical examination, clinical laboratory tests, vital sign measurements, and 12-lead electrocardiogram (ECG) at Screening and at upon admission to the Clinical Research Unit (CRU) and prior to administration of study intervention on Day 1.
5. Female study participants must not be a woman of childbearing potential and must either be postmenopausal (defined as no menses for 12 months without an alternative medical cause; follicle-stimulating hormone (FSH) to be tested for confirmation at Screening) or premenopausal with 1 of the following documented: hysterectomy, tubal ligation, bilateral salpingectomy, or bilateral oophorectomy.
6. Male study participants must agree to use contraception during the treatment period and for at least 3 months after the last dose of study intervention.

Exclusion Criteria:

1. Considered by the investigator or subinvestigator (suitably qualified) to be ineligible for the study due to a history of or current condition of significant metabolic or endocrine, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal (GI), urological, immunological, neurological, or psychiatric disorders with clinical manifestations.
2. History or presence of cancer in last 5 years except for non-melanoma skin cancers.
3. Risk factors for:

   1. Torsades de Pointes (eg, heart failure, cardiomyopathy, or family history of Long QT Syndrome or Brugada Syndrome)
   2. Unexplained syncope, sick sinus syndrome, second- or third-degree atrioventricular (AV) block, myocardial infarction, pulmonary congestion, cardiac arrhythmia, angina, prolonged QT interval, or conduction abnormalities
4. History of GI surgery or disease including, but not limited to, gastric band/gastric resection and/or intestinal resection and/or duodenal disease (ie, celiac disease) that may result in clinically significant malabsorption (except for an appendectomy).
5. History of hypersensitivity or severe side effects induced by a drug.
6. Any condition requiring medication and/or other treatment, such as dietary restriction and physical therapy.
7. History of significant multiple and/or severe allergic symptoms including food allergy (NOTE: Study participants with seasonal allergies may participate unless they have ongoing symptoms).
8. Used drugs or substances known to be inducers or inhibitors of cytochrome P450 enzymes and/or P-glycoprotein within 28 days prior to admission to the CRU.
9. Used prescription or over-the-counter (OTC) drugs, antacids, proton pump inhibitors, H2 antagonists, Chinese herbal medicines, oral cannabidiol, vitamins, minerals, herbal, and dietary supplements within 14 days prior to admission to the CRU.
10. Refuses to abstain from ingesting caffeine- or xanthine-containing products/medications (eg, coffee, tea, cola drinks, other caffeinated beverages, or chocolate) from 24 hours prior to admission to the CRU or refuses to refrain from consuming such products throughout the study (including Follow-up period).
11. Consumed alcohol or used alcohol-containing products within 72 hours prior to admission to the CRU or refuses to refrain from consuming such products throughout the study (including Follow-up period).
12. History of recreational drug use in the previous 6 months, or has a history of problematic alcohol use (defined as study participants who regularly consume excessive amounts of alcohol, defined as > 3 glasses of alcoholic beverages per day (1 glass is approximately equivalent to: beer [284 mL/10 ounces (oz.)], wine [125 mL/4 oz.] or distilled spirits [25 mL/1 oz.]).
13. A positive drug or alcohol screen at the Screening visit or upon admission to the CRU.
14. Used tobacco- or nicotine-containing products (including cigarette, pipe, cigar, chewing, nicotine patch, nicotine gum, or Vaping product) within 6 months prior to admission to the CRU or refuses to refrain from using tobacco- or nicotine-containing products throughout the study (including Follow-up period).
15. Consumed grapefruit, grapefruit juice, Seville orange juice, orange juice, apple juice, vegetables from the mustard green family (eg, kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard greens), or charbroiled meats within 7 days prior to admission to the CRU or refuses to refrain from consuming such products throughout the study (including Follow-up period).
16. A corrected QT (QTc) interval of > 450 msec for males and > 470 msec for females (Fridericia's method) at the Screening visit or upon admission to the CRU.
17. Systolic blood pressure is outside the range of 90 to 140 mm Hg, diastolic blood pressure is outside the range of 50 to 90 mm Hg, or pulse rate is outside the range of 40 to 100 beats per minute (bpm) or considered ineligible by the investigator or subinvestigator at the Screening visit or upon admission to the CRU.
18. Total bilirubin, alanine aminotransferase (ALT), or aspartate aminotransferase (AST) values are greater than the upper limit of normal (ULN), or estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73 m² at Screening or upon admission to the CRU.
19. A positive serological test for untreated syphilis, positive hepatitis B surface antigen, positive hepatitis C virus antibody, or positive human immunodeficiency virus (HIV) antigen/antibody result at the Screening visit.
20. Participated in any other investigational trials or has been exposed to other investigational drugs within 28 days or 5 half-lives of the previously administered investigational drug (date derived from last study procedure [blood collection or dosing] of previous trial), whichever is longer, prior to admission to the CRU.
21. Previously received S-648414.
22. Poor venous access.
23. Donated blood or had significant blood loss within 56 days of study admission to the CRU or donated plasma within 7 days prior to until admission to the CRU.
24. Considered inappropriate for participation in the study for any reason by the investigator or subinvestigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (2):
- PPD Ph 1 Clinical Research Unit, Austin, Texas, United States
- P-One Clinic, Hachiōji, Toyko, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of Part 1 (single ascending dose [SAD], food effect, and effects on electrocardiogram [ECG] parameters), Part 2 (multiple ascending dose [MAD] and drug-drug interaction with midazolam, a CYP3A substrate), and Part 3 (the effect of S-648414 on the pharmacokinetics (PK) of dolutegravir and the effect of dolutegravir on the PK of S-648414).
  Parts 1 and 2 were conducted at a single site in the United States, and Part 3 was conducted at a single site in Japan.
Pre-assignment Details: In Part 1 healthy participants were sequentially assigned to 1 of 6 ascending dose groups; within each dose group participants were randomized in a 3:1 ratio (4:1 in the 100 mg dose group) to receive S-648414 or placebo.
  In Part 2 healthy participants were assigned to 1 of 2 dose groups with 8 study participants randomized to receive S-648414 and 2 study participants receiving placebo per group.
  In Part 3 healthy participants were enrolled in 1 of 2 dose groups.
Groups:
- Part 1: Placebo: Participants received a single oral dose of matching placebo to S-648414 in a fasted state on Day 1. Two participants assigned to the 100 mg dose cohort also received a single oral dose of matching placebo in a fed state (after a high-fat meal) on Day 14.
- Part 2: Placebo + Midazolam: Participants received matching placebo to S-648414 once a day on Days 1 to 14 and a single oral dose of 5 mg midazolam alone on Day -2 and co-administered with the placebo dose on Day 14.
Period: Overall Study
Arm/Group | Part 1: Placebo | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414 | Part 2: Placebo + Midazolam | Part 2: 50 mg S-648414 + Midazolam | Part 2: 30 mg S-648414 + Midazolam | Part 3: 100 mg S-648414 + Dolutegravir | Part 3: 200 mg S-648414 + Dolutegravir
Started | 12 | 6 | 6 | 8 | 6 | 6 | 6 | 4 | 8 | 8 | 14 | 14
Completed | 12 | 6 | 6 | 8 | 6 | 6 | 6 | 2 | 7 | 8 | 14 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414 | Part 2: Placebo + Midazolam | Part 2: 50 mg S-648414 + Midazolam | Part 2: 30 mg S-648414 + Midazolam | Part 3: 100 mg S-648414 + Dolutegravir | Part 3: 200 mg S-648414 + Dolutegravir | Total
Number analyzed (Participants) | 12 | 6 | 6 | 8 | 6 | 6 | 6 | 4 | 8 | 8 | 14 | 14 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age data are reported separately for each part of the study.
  years
    Part 1: number analyzed (Participants) | 12 | 6 | 6 | 8 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 50
    Part 1 | 33.3 (8.53) | 38.0 (10.55) | 40.3 (8.98) | 35.5 (7.80) | 28.5 (5.68) | 32.5 (14.87) | 36.5 (11.22) |  |  |  |  |  | 34.8 (9.74)
    Part 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 8 | 8 | 0 | 0 | 20
    Part 2 |  |  |  |  |  |  |  | 36.0 (10.03) | 37.3 (9.97) | 34.4 (7.03) |  |  | 35.9 (8.51)
    Part 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 14 | 28
    Part 3 |  |  |  |  |  |  |  |  |  |  | 35.4 (6.70) | 34.9 (6.32) | 35.1 (6.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 2 | 1 | 0 | 0 | 10
  Male | 12 | 5 | 5 | 7 | 6 | 4 | 5 | 3 | 6 | 7 | 14 | 14 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 3 | 4 | 1 | 2 | 3 | 0 | 3 | 3 | 2 | 0 | 27
  Not Hispanic or Latino | 7 | 5 | 3 | 4 | 5 | 4 | 3 | 4 | 5 | 5 | 12 | 14 | 71
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 5 | 3 | 2 | 3 | 4 | 2 | 2 | 2 | 3 | 5 | 2 | 6 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 3 | 4 | 5 | 2 | 4 | 4 | 2 | 5 | 3 | 12 | 8 | 58
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE is any event not present before exposure to study drug or any event already present that worsens after exposure to study drug.
  A serious adverse event is any untoward medical occurrence that resulted in death, was life-threatening, required or prolonged inpatient hospitalization, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect, or other event that may have jeopardized the participant or required intervention to prevent one of the outcomes above.
  The investigator assessed the intensity of each AE according to the following:
  Grade 1 (Mild): No or minimal interference with usual activities.
  Grade 2 (Moderate): More than minimal interference with usual activities, intervention indicated.
  Grade 3 (Severe): Inability to perform usual activities, intervention or hospitalization indicated.
  Grade 4 (Potentially life-threatening): Inability to perform self-care, intervention indicated to prevent permanent impairment, disability, or death.
Time Frame: From dosing on Day 1 or Day 14 up to 10 days post dose
Population: The safety analysis population included all participants randomly assigned to study intervention who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Placebo - Fasted: Participants received a single oral dose of matching placebo to S-648414 in a fasted state on Day 1.
- Part 1: Placebo - Fed: Participants received a single dose of matching placebo to S-648414 in a fed state (after a high-fat meal) on Day 14.
- Part 1: 100 mg S-648414 Fasted: Participants received a single oral dose of 100 mg S-648414 in a fasted state on Day 1.
- Part 1: 100 mg S-648414 Fed: Participants received a single dose of 100 mg S-648414 in a fed state (after a high-fat meal) on Day 14.
Arm/Group | Part 1: Placebo - Fasted | Part 1: Placebo - Fed | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 Fasted | Part 1: 100 mg S-648414 Fed | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 12 | 2 | 6 | 6 | 8 | 8 | 6 | 6 | 6
Participants
  Any treatment-emergent adverse event (TEAE) | 2 | 0 | 0 | 1 | 2 | 2 | 1 | 1 | 2
  Any treatment-related TEAE | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Any TEAE with severity Grade 2 to 4 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Any TEAE with severity Grade 3 to 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any gastrointestinal AEs | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Any ocular AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Serious adverse events (SAEs) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any treatment-related SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any TEAE leading to study discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any TEAE leading to study drug discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part 2: Number of Participants With Treatment-emergent Adverse Events
Description: as for outcome 1
Time Frame: From the first dose up to 10 days after end of dosing (25 days); A TEAE was summarized to a given treatment if the event onset/worsening occurred any time after the dose of that treatment and before the dose of the next treatment.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Midazolam (Day -2): Participants received a single oral dose of 5 mg midazolam on Day -2.
- Part 2: Placebo (Days 1-13): Participants received matching placebo to S-648414 orally once a day on Days 1 to 13.
- Part 2: 50 mg S-648414 (Days 1-13): Participants received 50 mg S-648414 orally once a day on Days 1 to 13.
- Part 2: 30 mg S-648414 (Days 1-13): Participants received 30 mg S-648414 orally once a day on Days 1 to 13.
- Part 2: Placebo + Midazolam (Day 14): Participants received matching placebo to S-648414 and a single oral dose of 5 mg midazolam on Day 14.
- Part 2: 50 mg S-648414 + Midazolam (Day 14): Participants received 50 mg S-648414 and a single oral dose of 5 mg midazolam on Day 14.
- Part 2: 30 mg S-648414 + Midazolam (Day 14): Participants received 30 mg S-648414 and a single oral dose of 5 mg midazolam on Day 14.
Arm/Group | Part 2: Midazolam (Day -2) | Part 2: Placebo (Days 1-13) | Part 2: 50 mg S-648414 (Days 1-13) | Part 2: 30 mg S-648414 (Days 1-13) | Part 2: Placebo + Midazolam (Day 14) | Part 2: 50 mg S-648414 + Midazolam (Day 14) | Part 2: 30 mg S-648414 + Midazolam (Day 14)
Number analyzed (Participants) | 20 | 4 | 8 | 8 | 2 | 7 | 8
Participants
  Any TEAE | 0 | 2 | 2 | 3 | 0 | 1 | 1
  Any treatment-related TEAE | 0 | 2 | 2 | 2 | 0 | 1 | 0
  Any TEAE with severity Grade 2 to 4 | 0 | 2 | 2 | 1 | 0 | 0 | 0
  Any TEAE with severity Grade 3 to 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any gastrointestinal AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any ocular AEs | 0 | 1 | 0 | 2 | 0 | 0 | 0
  Any serious adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any treatment-related SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any TEAE leading to study discontinuation | 0 | 2 | 1 | 0 | 0 | 0 | 0
  Any TEAE leading to study drug discontinuation | 0 | 2 | 1 | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Part 3: Number of Participants With Treatment-emergent Adverse Events
Description: as for outcome 1
Time Frame: From the first dose up to Day 36; A TEAE was summarized to a given treatment if the event onset/worsening occurred any time after the dose of that treatment and before the dose of the next treatment.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Part 3: Dolutegravir (100 mg S-648414 Group): Participants assigned to the 100 mg S-648414 dose group received 50 mg dolutegravir orally once a day on Days 1 to 7.
- Part 3: 100 mg S-648414: Participants received 100 mg S-648414 orally once a day on Days 15 to 21.
- Part 3: 100 mg S-648414 + Dolutegravir: Participants received 50 mg dolutegravir co-administered with 100 mg S-648414 orally once a day on Days 22 to 28.
- Part 3: Dolutegravir (200 mg S-648414 Group): Participants assigned to the 200 mg S-648414 dose group received 50 mg dolutegravir once a day on Days 1 to 7.
- Part 3: 200 mg S-648414: Participants received 200 mg S-648414 orally once a day on Days 15 to 21.
- Part 3: 200 mg S-648414 + Dolutegravir: Participants received 50 mg dolutegravir once a day co-administered with 200 mg S-648414 orally once a day on Days 22 to 28.
Arm/Group | Part 3: Dolutegravir (100 mg S-648414 Group) | Part 3: 100 mg S-648414 | Part 3: 100 mg S-648414 + Dolutegravir | Part 3: Dolutegravir (200 mg S-648414 Group) | Part 3: 200 mg S-648414 | Part 3: 200 mg S-648414 + Dolutegravir
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
Participants
  Any TEAE | 3 | 3 | 4 | 2 | 5 | 2
  Any treatment-related TEAE | 0 | 0 | 0 | 0 | 2 | 1
  Any TEAE with severity Grade 2 to 4 | 2 | 2 | 2 | 2 | 3 | 1
  Any TEAE with severity Grade 3 to 4 | 0 | 0 | 0 | 0 | 0 | 0
  Any gastrointestinal AEs | 0 | 0 | 0 | 0 | 0 | 1
  Any ocular AEs | 0 | 0 | 0 | 0 | 2 | 0
  Any serious adverse events | 0 | 0 | 0 | 0 | 0 | 0
  Any treatment-related SAE | 0 | 0 | 0 | 0 | 0 | 0
  Any TEAE leading to study discontinuation | 0 | 0 | 0 | 0 | 0 | 0
  Any TEAE leading to study drug discontinuation | 0 | 0 | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part 3: Maximum Plasma Concentration (Cmax) of S-648414
Description: The effect of dolutegravir on the pharmacokinetics (PK) of S-648414 was assessed after administration of multiple oral doses of S-648414 alone (Day 21) and after administration of multiple oral doses of S-648414 co-administered with dolutegravir (Day 28).
Time Frame: Day 21 predose (0 hours), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8 and 12 hours postdose. Day 28 predose (0 hours), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours postdose.
Population: The PK parameter population includes all study participants with at least 1 PK parameter estimated appropriately.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 3: 100 mg S-648414 | Part 3: 100 mg S-648414 + Dolutegravir | Part 3: 200 mg S-648414 | Part 3: 200 mg S-648414 + Dolutegravir
Number analyzed (Participants) | 14 | 14 | 14 | 14
ng/mL | 2740 (20.3) | 2720 (21.3) | 5150 (14.1) | 5020 (15.3)
Statistical Analysis 1: Comparison: Part 3: 100 mg S-648414 vs Part 3: 100 mg S-648414 + Dolutegravir; The effect of dolutegravir on the PK of S-648414 was assessed by analysis of variance (ANOVA) fit with a linear mixed effect model with the natural log (ln)-transformed Cmax as the dependent variable, treatment as fixed effect, and participant as random effect. The difference and 90% confidence interval (CI) between the ln-transformed Cmax of S-648414 + dolutegravir and S-648414 alone were estimated then back-transformed to obtain the corresponding geometric least squares mean ratio and 90% CI; Test type: Other — The drug interaction was assessed by whether the 90% CIs for the geometric least squares mean ratio of Cmax, Cτ, and AUC0-τ of S-648414 were completely contained within the range of 0.8000 to 1.2500; Geometric Least Squares Mean Ratio = 0.9913, 90% CI 2-sided [0.9232 to 1.0645] — Ratio = S-648414 + Dolutegravir / S-648414
Statistical Analysis 2: Comparison: Part 3: 200 mg S-648414 vs Part 3: 200 mg S-648414 + Dolutegravir; The effect of dolutegravir on the PK of S-648414 was assessed by an ANOVA fitted with a linear mixed effect model with the natural log-transformed Cmax as the dependent variable, treatment as fixed effect, and participant as random effect. The difference and 90% CI between the ln-transformed Cmax of S-648414 + dolutegravir and S-648414 alone were estimated then back-transformed to obtain the corresponding geometric least squares mean ratio and 90% CI; Test type: Other — [test comment as in outcome 4, analysis 1]; Geometric Least Squares Mean Ratio = 0.9754, 90% CI 2-sided [0.8916 to 1.0671] — Ratio = S-648414 + Dolutegravir / S-648414

5. Primary Outcome: Part 3: Time to Maximum Plasma Concentration (Tmax) of S-648414
Description: as for outcome 4
Time Frame: as for outcome 4
Population: The PK parameter population
Measure: Median (Full Range); unit: hours
Arm/Group | Part 3: 100 mg S-648414 | Part 3: 100 mg S-648414 + Dolutegravir | Part 3: 200 mg S-648414 | Part 3: 200 mg S-648414 + Dolutegravir
Number analyzed (Participants) | 14 | 14 | 14 | 14
hours | 2.00 [1.00 to 4.00] | 2.25 [1.00 to 5.00] | 2.50 [1.00 to 4.00] | 2.25 [1.00 to 5.00]

6. Primary Outcome: Part 3: Plasma Concentration of S-648414 at the End of the Dosing Interval τ (Cτ)
Description: as for outcome 4
Time Frame: Day 22 and Day 29 (24 hours post-dosing on Days 21 and 28)
Population: The PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 3: 100 mg S-648414 | Part 3: 100 mg S-648414 + Dolutegravir | Part 3: 200 mg S-648414 | Part 3: 200 mg S-648414 + Dolutegravir
Number analyzed (Participants) | 14 | 14 | 14 | 14
ng/mL | 1210 (27.7) | 1250 (16.3) | 2590 (16.5) | 2360 (14.5)
Statistical Analysis 1: Comparison: Part 3: 100 mg S-648414 vs Part 3: 100 mg S-648414 + Dolutegravir; The effect of dolutegravir on the PK of S-648414 was assessed using an ANOVA fitted with a linear mixed effect model with the natural log-transformed Cτ as the dependent variable, treatment as a fixed effect, and participant as a random effect. The difference and 90% CI between the ln-transformed Cτ of S-648414 + dolutegravir and S-648414 alone were estimated then back-transformed to obtain the corresponding geometric least squares mean ratio and 90% CI; Test type: Other — [test comment as in outcome 4, analysis 1]; Geometric Least Squares Mean Ratio = 1.0353, 90% CI 2-sided [0.9421 to 1.1377] — Ratio = S-648414 + Dolutegravir / S-648414
Statistical Analysis 2: Comparison: Part 3: 200 mg S-648414 vs Part 3: 200 mg S-648414 + Dolutegravir; [analysis description as in outcome 6, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; Geometric Least Squares Mean Ratio = 0.9096, 90% CI 2-sided [0.8791 to 0.9411] — Ratio = S-648414 + Dolutegravir / S-648414

7. Primary Outcome: Part 3: Area Under the Concentration-time Curve Over the Dosing Interval τ (AUC0-τ) for S-648414
Description: The effect of dolutegravir on the pharmacokinetics (PK) of S-648414 was assessed after administration of multiple oral doses of S-648414 alone (Day 21) and after administration of multiple oral doses of S-648414 co-administered with dolutegravir (Day 28).
  Area under the concentration-time curve over the dosing interval τ (24 hours) was calculated by the linear up/log down trapezoidal method.
Time Frame: as for outcome 4
Population: The PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 3: 100 mg S-648414 | Part 3: 100 mg S-648414 + Dolutegravir | Part 3: 200 mg S-648414 | Part 3: 200 mg S-648414 + Dolutegravir
Number analyzed (Participants) | 14 | 14 | 14 | 14
ng*hr/mL | 40800 (17.6) | 41080 (15.4) | 81010 (11.4) | 79820 (12.5)
Statistical Analysis 1: Comparison: Part 3: 100 mg S-648414 vs Part 3: 100 mg S-648414 + Dolutegravir; The effect of dolutegravir on the PK of S-648414 was assessed using an ANOVA fitted with a linear mixed effect model with the natural log-transformed AUC0-τ as the dependent variable, treatment as a fixed effect, and participant as a random effect. The difference and 90% CI between the ln-transformed AUC0-τ of S-648414 + dolutegravir and S-648414 alone were estimated then back-transformed to obtain the corresponding geometric least squares mean ratio and 90% CI; Test type: Other — [test comment as in outcome 4, analysis 1]; Geometric Least Squares Mean Ratio = 1.0071, 90% CI 2-sided [0.9679 to 1.0479] — Ratio = S-648414 + Dolutegravir / S-648414
Statistical Analysis 2: Comparison: Part 3: 200 mg S-648414 vs Part 3: 200 mg S-648414 + Dolutegravir; [analysis description as in outcome 7, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; Geometric Least Squares Mean Ratio = 0.9852, 90% CI 2-sided [0.9605 to 1.0105] — Ratio = S-648414 + Dolutegravir / S-648414

8. Primary Outcome: Part 3: Apparent Total Clearance (CL/F) of S-648414
Description: The effect of dolutegravir on the pharmacokinetics (PK) of S-648414 was assessed after administration of multiple oral doses of S-648414 alone (Day 21) and after administration of multiple oral doses of S-648414 co-administered with dolutegravir (Day 28).
  Apparent total clearance was calculated as CL/F = Dose/AUC0-τ
Time Frame: as for outcome 4
Population: The PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Part 3: 100 mg S-648414 | Part 3: 100 mg S-648414 + Dolutegravir | Part 3: 200 mg S-648414 | Part 3: 200 mg S-648414 + Dolutegravir
Number analyzed (Participants) | 14 | 14 | 14 | 14
L/hr | 2.45 (17.6) | 2.43 (15.4) | 2.47 (11.4) | 2.51 (12.5)

9. Primary Outcome: Part 3: Maximum Plasma Concentration (Cmax) of Dolutegravir
Description: The effect of S-648414 on the PK of dolutegravir was assessed after administration of multiple oral doses of dolutegravir alone and after administration of multiple oral doses of S-648414 co-administered with dolutegravir.
Time Frame: Day 7 and Day 28 predose (0 hours), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 and 24 hours postdose.
Population: The PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 3: Dolutegravir (100 mg S-648414 Group) | Part 3: 100 mg S-648414 + Dolutegravir | Part 3: Dolutegravir (200 mg S-648414 Group) | Part 3: 200 mg S-648414 + Dolutegravir
Number analyzed (Participants) | 14 | 14 | 14 | 14
ng/mL | 4910 (15.9) | 5800 (12.2) | 4720 (19.6) | 4950 (15.9)
Statistical Analysis 1: Comparison: Part 3: Dolutegravir (100 mg S-648414 Group) vs Part 3: 100 mg S-648414 + Dolutegravir; The effect of S-648414 on the plasma PK of dolutegravir was assessed using an ANOVA fitted with a linear mixed effect model with the natural log-transformed Cmax as the dependent variable, treatment as a fixed effect, and participant as a random effect. The difference and 90% CI between the ln-transformed Cmax of dolutegravir plus S-648414 and dolutegravir alone was estimated then back-transformed to obtain the corresponding geometric least squares mean ratio and 90% CI; Test type: Other — The drug interaction was assessed by whether the 90% CIs for the geometric least squares mean ratio of Cmax, Cτ, and AUC0-τ of dolutegravir were completely contained within the range of 0.8000 to 1.2500; Geometric Least Squares Mean Ratio = 1.1806, 90% CI 2-sided [1.1171 to 1.2477] — Ratio = S-648414 + Dolutegravir / Dolutegravir
Statistical Analysis 2: Comparison: Part 3: Dolutegravir (200 mg S-648414 Group) vs Part 3: 200 mg S-648414 + Dolutegravir; [analysis description as in outcome 9, analysis 1]; Test type: Other — [test comment as in outcome 9, analysis 1]; Geometric Least Squares Mean Ratio = 1.0480, 90% CI 2-sided [0.9656 to 1.1373] — Ratio = S-648414 + Dolutegravir / Dolutegravir

10. Primary Outcome: Part 3: Time to Maximum Plasma Concentration (Tmax) of Dolutegravir
Description: as for outcome 9
Time Frame: Day 7 and Day 28 predose (0 hours), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 and 24 hours postdose.
Population: The PK parameter population
Measure: Median (Full Range); unit: hours
Arm/Group | Part 3: Dolutegravir (100 mg S-648414 Group) | Part 3: 100 mg S-648414 + Dolutegravir | Part 3: Dolutegravir (200 mg S-648414 Group) | Part 3: 200 mg S-648414 + Dolutegravir
Number analyzed (Participants) | 14 | 14 | 14 | 14
hours | 3.50 [1.50 to 4.00] | 2.75 [1.00 to 4.00] | 3.50 [1.00 to 5.00] | 4.00 [1.50 to 5.00]

11. Primary Outcome: Part 3: Plasma Concentration of Dolutegravir at the End of the Dosing Interval τ (Cτ)
Description: as for outcome 9
Time Frame: Day 8 and Day 29 (24 hours post-dosing on Day 7 and Day 28).
Population: The PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 3: Dolutegravir (100 mg S-648414 Group) | Part 3: 100 mg S-648414 + Dolutegravir | Part 3: Dolutegravir (200 mg S-648414 Group) | Part 3: 200 mg S-648414 + Dolutegravir
Number analyzed (Participants) | 14 | 14 | 14 | 14
ng/mL | 1980 (23.1) | 2660 (17.6) | 1850 (25.7) | 2000 (23.9)
Statistical Analysis 1: Comparison: Part 3: Dolutegravir (100 mg S-648414 Group) vs Part 3: 100 mg S-648414 + Dolutegravir; The effect of S-648414 on the plasma PK of dolutegravir was assessed using an ANOVA fitted with a linear mixed effect model with the natural log-transformed Cτ as the dependent variable, treatment as a fixed effect, and participant as a random effect. The difference and 90% CI between the ln-transformed Cτ of dolutegravir plus S-648414 and dolutegravir alone was estimated then back-transformed to obtain the corresponding geometric least squares mean ratio and 90% CI; Test type: Other — [test comment as in outcome 9, analysis 1]; Geometric Least Squares Mean Ratio = 1.3445, 90% CI 2-sided [1.2352 to 1.4636] — Ratio = S-648414 + Dolutegravir / Dolutegravir
Statistical Analysis 2: Comparison: Part 3: Dolutegravir (200 mg S-648414 Group) vs Part 3: 200 mg S-648414 + Dolutegravir; [analysis description as in outcome 11, analysis 1]; Test type: Other — [test comment as in outcome 9, analysis 1]; Geometric Least Squares Mean Ratio = 1.0769, 90% CI 2-sided [1.0137 to 1.1441] — Ratio = S-648414 + Dolutegravir / Dolutegravir

12. Primary Outcome: Part 3: Area Under the Concentration-time Curve Over the Dosing Interval τ (AUC0-τ) for Dolutegravir
Description: The effect of S-648414 on the PK of dolutegravir was assessed after administration of multiple oral doses of dolutegravir alone and after administration of multiple oral doses of S-648414 co-administered with dolutegravir.
  Area under the concentration-time curve over the dosing interval τ (24 hours) was calculated by the linear up/log down trapezoidal method.
Time Frame: Day 7 and Day 28 predose (0 hours), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 and 24 hours postdose.
Population: The PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 3: Dolutegravir (100 mg S-648414 Group) | Part 3: 100 mg S-648414 + Dolutegravir | Part 3: Dolutegravir (200 mg S-648414 Group) | Part 3: 200 mg S-648414 + Dolutegravir
Number analyzed (Participants) | 14 | 14 | 14 | 14
ng*hr/mL | 74790 (19.7) | 89290 (13.4) | 69850 (20.1) | 73210 (17.6)
Statistical Analysis 1: Comparison: Part 3: Dolutegravir (100 mg S-648414 Group) vs Part 3: 100 mg S-648414 + Dolutegravir; The effect of S-648414 on the plasma PK of dolutegravir was assessed using an ANOVA fitted with a linear mixed effect model with the natural log-transformed AUC0-τ as the dependent variable, treatment as a fixed effect, and participant as a random effect. The difference and 90% CI between the ln-transformed AUC0-τ of dolutegravir plus S-648414 and dolutegravir alone was estimated then back-transformed to obtain the corresponding geometric least squares mean ratio and 90% CI; Test type: Other — [test comment as in outcome 9, analysis 1]; Geometric Least Squares Mean Ratio = 1.1939, 90% CI 2-sided [1.1176 to 1.2754] — Ratio = S-648414 + Dolutegravir / Dolutegravir
Statistical Analysis 2: Comparison: Part 3: Dolutegravir (200 mg S-648414 Group) vs Part 3: 200 mg S-648414 + Dolutegravir; [analysis description as in outcome 12, analysis 1]; Test type: Other — [test comment as in outcome 9, analysis 1]; Geometric Least Squares Mean Ratio = 1.0482, 90% CI 2-sided [0.9881 to 1.1119] — Ratio = S-648414 + Dolutegravir / Dolutegravir

13. Primary Outcome: Part 3: Apparent Total Clearance (CL/F) of Dolutegravir
Description: The effect of S-648414 on the PK of dolutegravir was assessed after administration of multiple oral doses of dolutegravir alone and after administration of multiple oral doses of S-648414 co-administered with dolutegravir.
  Apparent total clearance calculated as CL/F =Dose/AUC0-τ
Time Frame: Day 7 and Day 28 predose (0 hours), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12 and 24 hours postdose.
Population: The PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Part 3: Dolutegravir (100 mg S-648414 Group) | Part 3: 100 mg S-648414 + Dolutegravir | Part 3: Dolutegravir (200 mg S-648414 Group) | Part 3: 200 mg S-648414 + Dolutegravir
Number analyzed (Participants) | 14 | 14 | 14 | 14
L/hr | 0.669 (19.7) | 0.560 (13.4) | 0.716 (20.1) | 0.683 (17.6)

14. Secondary Outcome: Part 1: Maximum Plasma Concentration (Cmax) of S-648414
Time Frame: Day 1 and Day 14 (for participants in the 100 mg dose group only) predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72 and 96 hours postdose.
Population: The PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 Fasted | Part 1: 100 mg S-648414 Fed | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 6 | 6 | 6
ng/mL | 151 (22.8) | 498 (17.7) | 1620 (13.1) | 1430 (18.0) | 3820 (25.7) | 9260 (31.9) | 12700 (26.3)
Statistical Analysis 1: Comparison: Part 1: 10 mg S-648414 vs Part 1: 30 mg S-648414 vs Part 1: 100 mg S-648414 Fasted vs Part 1: 250 mg S-648414 vs Part 1: 500 mg S-648414 vs Part 1: 1000 mg S-648414; The dose proportionality of plasma PK parameters of S-648414 was examined for all fasted groups in Part 1 using the power model. The power model assumes a linear relationship between the ln-transformed parameter and ln-transformed dose where ln(Cmax) = Intercept + Slope × ln(Dose) + Random error; Test type: Other; Slope = 0.9857, 95% CI 2-sided [0.9341 to 1.0373]
Statistical Analysis 2: Comparison: Part 1: 100 mg S-648414 Fasted vs Part 1: 100 mg S-648414 Fed; The effect of food on the plasma PK of S-648414 was examined after a single dose of 100 mg S-648414 in the fed state and fasted state using an ANOVA fitted with a linear mixed effect model with ln-transformed Cmax as the dependent variable, treatment as a fixed effect, and participant as random effect. The difference and 90% CI between the fed and fasted state ln-transformed Cmax were estimated, then back-transformed to obtain the corresponding geometric least squares mean ratio and 90% CI; Test type: Other; Geometric Least Squares Mean Ratio = 0.8786, 90% CI 2-sided [0.7705 to 1.0019] — Ratio = Fed / Fasted

15. Secondary Outcome: Part 1: Time to Maximum Plasma Concentration (Tmax) of S-648414
Time Frame: as for outcome 14
Population: The PK parameter population
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 Fasted | Part 1: 100 mg S-648414 Fed | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 6 | 6 | 6
hours | 1.00 [1.00 to 1.50] | 1.00 [1.00 to 2.00] | 1.25 [1.00 to 1.50] | 3.00 [2.00 to 6.00] | 1.50 [1.00 to 2.00] | 1.50 [1.03 to 4.00] | 1.75 [1.50 to 3.00]

16. Secondary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration After Dosing (AUC0-last) of S-648414
Description: Area under the concentration-time curve from time zero to the time of the last quantifiable concentration after dosing, calculated by the linear trapezoidal method when concentrations are increasing and by the logarithmic trapezoidal method when concentrations are decreasing (linear up/log down trapezoidal method).
Time Frame: as for outcome 14
Population: The PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 Fasted | Part 1: 100 mg S-648414 Fed | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 6 | 6 | 6
ng*hr/mL | 3431 (18.1) | 10610 (19.3) | 36370 (9.2) | 34910 (14.2) | 89330 (20.2) | 215300 (27.1) | 359300 (23.3)
Statistical Analysis 1: Comparison: Part 1: 10 mg S-648414 vs Part 1: 30 mg S-648414 vs Part 1: 100 mg S-648414 Fasted vs Part 1: 250 mg S-648414 vs Part 1: 500 mg S-648414 vs Part 1: 1000 mg S-648414; The dose proportionality of plasma PK parameters of S-648414 was examined for all fasted groups in Part 1 using the power model. The power model assumes a linear relationship between the ln-transformed parameter and ln-transformed dose where ln(AUC0-last) = Intercept + Slope × ln(Dose) + Random error; Test type: Other; Slope = 1.0252, 95% CI 2-sided [0.9840 to 1.0665]
Statistical Analysis 2: Comparison: Part 1: 100 mg S-648414 Fasted vs Part 1: 100 mg S-648414 Fed; The effect of food on the plasma PK of S-648414 was examined after a single dose of 100 mg S-648414 in the fed and fasted state using an ANOVA fitted with a linear mixed effect model, with ln-transformed AUC0-last as the dependent variable, treatment as a fixed effect, and participant as random effect. The difference and 90% CI between the fed and fasted state ln-transformed AUC0-last were estimated, then back-transformed to obtain the corresponding geometric least squares mean ratio and 90% CI; Test type: Other; Geometric Least Squares Mean Ratio = 0.9598, 90% CI 2-sided [0.8585 to 1.0730] — Ratio = Fed / Fasted

17. Secondary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of S-648414
Description: Area under the concentration-time curve extrapolated from time zero to infinity defined as AUC0-last + (Clast/λz), where Clast is the last measurable plasma concentration and λz is the plasma terminal elimination rate constant.
Time Frame: as for outcome 14
Population: The PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 Fasted | Part 1: 100 mg S-648414 Fed | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 6 | 6 | 6
ng*hr/mL | 3620 (17.5) | 11040 (19.6) | 38300 (10.9) | 36940 (14.4) | 95510 (21.0) | 226600 (26.5) | 382000 (23.6)
Statistical Analysis 1: Comparison: Part 1: 10 mg S-648414 vs Part 1: 30 mg S-648414 vs Part 1: 100 mg S-648414 Fasted vs Part 1: 250 mg S-648414 vs Part 1: 500 mg S-648414 vs Part 1: 1000 mg S-648414; The dose proportionality of plasma PK parameters of S-648414 was examined for all fasted groups in Part 1 using the power model. The power model assumes a linear relationship between the ln-transformed parameter and ln-transformed dose where ln(AUC0-inf) = Intercept + Slope × ln(Dose) + Random error; Test type: Other; Slope = 1.0280, 95% CI 2-sided [0.9866 to 1.0695]
Statistical Analysis 2: Comparison: Part 1: 100 mg S-648414 Fasted vs Part 1: 100 mg S-648414 Fed; The effect of food on the plasma PK of S-648414 was examined after a single dose of 100 mg S-648414 in the fed and fasted state using an ANOVA fitted with a linear mixed effect model, with ln-transformed AUC0-inf as the dependent variable, treatment as a fixed effect, and participant as random effect. The difference and 90% CI between the fed and fasted state ln-transformed AUC0-inf were estimated, then back-transformed to obtain the corresponding geometric least squares mean ratio and 90% CI; Test type: Other; Geometric Least Squares Mean Ratio = 0.9646, 90% CI 2-sided [0.8643 to 1.0766] — Ratio = Fed / Fasted

18. Secondary Outcome: Part 1: Terminal Elimination Half-life (t1/2,z) of S-648414
Description: Terminal elimination half-life calculated as t1/2,z = (ln2)/λz, where λz is the terminal elimination rate constant.
Time Frame: as for outcome 14
Population: The PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 Fasted | Part 1: 100 mg S-648414 Fed | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 6 | 6 | 6
hours | 23.0 (5.0) | 20.7 (9.9) | 22.2 (16.0) | 22.8 (14.2) | 24.1 (12.1) | 22.2 (12.1) | 23.7 (14.2)
Statistical Analysis 1: Comparison: Part 1: 100 mg S-648414 Fasted vs Part 1: 100 mg S-648414 Fed; The effect of food on the plasma PK of S-648414 was examined after a single dose of 100 mg S-648414 in the fed and fasted state using an ANOVA fitted with a linear mixed effect model, with ln-transformed t1/2,z as the dependent variable, treatment as a fixed effect, and participant as random effect. The difference and 90% CI between the fed and fasted state ln-transformed t1/2,z were estimated, then back-transformed to obtain the corresponding geometric least squares mean ratio and 90% CI; Test type: Other; Geometric Least Squares Mean Ratio = 1.0272, 90% CI 2-sided [0.9949 to 1.0606] — Ratio = Fed / Fasted

19. Secondary Outcome: Part 1: Terminal Elimination Rate Constant (λz) of S-648414
Time Frame: as for outcome 14
Population: The PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 Fasted | Part 1: 100 mg S-648414 Fed | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 6 | 6 | 6
1/hour | 0.0301 (5.0) | 0.0336 (9.9) | 0.0313 (16.0) | 0.0305 (14.2) | 0.0288 (12.1) | 0.0312 (12.1) | 0.0293 (14.2)

20. Secondary Outcome: Part 1: Mean Residence Time (MRT) of S-648414
Description: Mean residence time, calculated as MRT = AUMC0-inf / AUC0-inf, where AUMC0-inf is the area under the first moment curve extrapolated to infinity.
Time Frame: as for outcome 14
Population: The PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 Fasted | Part 1: 100 mg S-648414 Fed | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 6 | 6 | 6
hours | 32.5 (4.3) | 29.2 (9.5) | 31.5 (16.1) | 33.8 (14.6) | 34.2 (12.6) | 32.6 (12.9) | 34.5 (13.3)

21. Secondary Outcome: Part 1: Apparent Total Clearance (CL/F) of S-648414
Description: Apparent total clearance estimated according to: CL/F = Dose / AUC0-inf.
Time Frame: as for outcome 14
Population: The PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 Fasted | Part 1: 100 mg S-648414 Fed | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 6 | 6 | 6
L/hr | 2.76 (17.5) | 2.72 (19.6) | 2.61 (10.9) | 2.71 (14.4) | 2.62 (21.0) | 2.21 (26.5) | 2.62 (23.6)

22. Secondary Outcome: Part 1: Apparent Volume of Distribution in the Terminal Elimination Phase (Vz/F) of S-648414
Description: Apparent volume of distribution in the terminal elimination phase was estimated according to: Vz /F = Dose / AUC0-inf / λz.
Time Frame: as for outcome 14
Population: The PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 Fasted | Part 1: 100 mg S-648414 Fed | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 6 | 6 | 6
liters | 91.7 (21.2) | 81.0 (21.2) | 83.5 (11.0) | 88.9 (19.5) | 91.0 (17.3) | 70.8 (31.7) | 89.3 (23.9)

23. Secondary Outcome: Part 1: Fraction of S-648414 Dose Excreted in Urine From 0 to 96 Hours Postdose (Feu0-96)
Description: The fraction of S-648414 dose excreted in urine from 0 to 96 hours postdose was calculated as:
  Cumulative amount of S-648414 excreted in urine from time zero to 96 hours postdose (Aeu0-96) / Dose × 100
Time Frame: Day 1 and Day 14 (for participants in the 100 mg dose group only) predose (-12 to 0 hours), 0 to 24 hours, 24 to 48 hours, 48 to 72 hours, and 72 to 96 hours postdose
Population: The PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent excreted
Arm/Group | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 Fasted | Part 1: 100 mg S-648414 Fed | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 6 | 6 | 6
percent excreted | 30.3 (22.6) | 25.5 (20.1) | 25.3 (19.2) | 25.1 (11.1) | 28.7 (19.8) | 31.5 (10.2) | 25.9 (27.3)

24. Secondary Outcome: Part 1: Renal Clearance (CLR) of S-648414
Description: Renal clearance was estimated according to: CLR = cumulative amount of S-648414 excreted in urine from time zero to 96 hours postdose (Aeu0-96) / area under the concentration-time curve from time zero to the time of the last quantifiable concentration after dosing (AUC0-last).
Time Frame: as for outcome 23
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 Fasted | Part 1: 100 mg S-648414 Fed | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 6 | 6 | 6
L/hr | 0.884 (11.6) | 0.721 (25.9) | 0.695 (17.5) | 0.720 (18.4) | 0.804 (10.3) | 0.732 (30.6) | 0.720 (24.3)

25. Secondary Outcome: Part 2: Maximum Plasma Concentration (Cmax) of S-648414 Following Single and Multiple-dose Administration
Time Frame: Day 1 predose (0 hours), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours postdose; Day 14 predose (0 hours), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, and 96 hours postdose.
Population: The PK parameter population with available data at each time point
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: 30 mg S-648414 + Midazolam | Part 2: 50 mg S-648414 + Midazolam
Number analyzed (Participants) | 8 | 8
ng/mL
  Day 1 | 411 (22.3) | 623 (19.2)
  Day 14: number analyzed (Participants) | 8 | 6
  Day 14 | 719 (13.2) | 1320 (20.2)
Statistical Analysis 1: Comparison: Part 2: 30 mg S-648414 + Midazolam vs Part 2: 50 mg S-648414 + Midazolam; The dose proportionality of plasma S-648414 Cmax after a single dose of S-648414 (Day 1) was assessed using an ANOVA model fitted to the ln-transformed Cmax, with dose group fitted as a fixed factor. The point estimates and 90% CIs were generated for the ratios of the 50 mg dose to 30 mg dose ln-transformed Cmax, then back-transformed to obtain the corresponding geometric least squares mean ratio and 90% CI; Test type: Other; Geometric Least Squares Mean Ratio = 1.5167, 90% CI 2-sided [1.2654 to 1.8180] — Ratio = 50 mg / 30 mg
Statistical Analysis 2: Comparison: Part 2: 30 mg S-648414 + Midazolam vs Part 2: 50 mg S-648414 + Midazolam; The dose proportionality of plasma S-648414 Cmax after multiple doses of S-648414 (Day 14) was assessed using an ANOVA model fitted to the ln-transformed Cmax, with dose group fitted as a fixed factor. The point estimates and 90% CIs were generated for the ratios of the 50 mg dose to 30 mg dose ln-transformed Cmax, then back-transformed to obtain the corresponding geometric least squares mean ratio and 90% CI; Test type: Other; Geometric Least Squares Mean Ratio = 1.8372, 90% CI 2-sided [1.5696 to 2.1506] — Ratio = 50 mg / 30 mg
Statistical Analysis 3: Comparison: Part 2: 30 mg S-648414 + Midazolam; The accumulation ratio of Cmax in the 30 mg dose group was calculated as the ratio of Day 14 to Day 1 using an ANOVA fitted with a linear mixed model with ln-transformed Cmax, Day as a fixed effect and participant as a random effect. The difference and 90% CI between the ln-transformed Cmax on Day 1 and Day 14 were estimated then back-transformed to obtain the corresponding geometric least squares mean ratio and 90% CI; Test type: Other; Geometric Least Squares Mean Ratio = 1.7489, 90% CI 2-sided [1.5250 to 2.0057] — Ratio = Day 14 / Day 1
Statistical Analysis 4: Comparison: Part 2: 50 mg S-648414 + Midazolam; The accumulation ratio of Cmax in the 50 mg dose group was calculated as the ratio of Day 14 to Day 1 using an ANOVA fitted with a linear mixed model with ln-transformed Cmax, Day as a fixed effect and participant as a random effect. The difference and 90% CI between the ln-transformed Cmax on Day 1 and Day 14 were estimated then back-transformed to obtain the corresponding geometric least squares mean ratio and 90% CI; Test type: Other; Geometric Least Squares Mean Ratio = 2.1453, 90% CI 2-sided [1.9741 to 2.3313] — Ratio = Day 14 / Day 1

26. Secondary Outcome: Part 2: Time to Maximum Plasma Concentration (Tmax) of S-648414 Following Single and Multiple-dose Administration
Time Frame: as for outcome 25
Population: The PK parameter population with available data at each time point
Measure: Median (Full Range); unit: hours
Arm/Group | Part 2: 30 mg S-648414 + Midazolam | Part 2: 50 mg S-648414 + Midazolam
Number analyzed (Participants) | 8 | 8
hours
  Day 1 | 3.02 [2.00 to 5.00] | 4.50 [2.50 to 5.00]
  Day 14: number analyzed (Participants) | 8 | 6
  Day 14 | 2.03 [1.50 to 5.12] | 1.25 [1.00 to 2.50]

27. Secondary Outcome: Part 2: Area Under the Concentration-time Curve Over the Dosing Interval τ (AUC0-τ) of S-648414 Following Single and Multiple-dose Administration
Description: Area under the concentration-time curve over the dosing interval (24 hours) on Day 1 and Day 14, calculated by the linear up/log down trapezoidal method.
Time Frame: Day 1 and day 14 predose (0 hours), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours postdose.
Population: The PK parameter population with available data at each time point
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 2: 30 mg S-648414 + Midazolam | Part 2: 50 mg S-648414 + Midazolam
Number analyzed (Participants) | 8 | 8
ng*hr/mL
  Day 1 | 5519 (15.9) | 8983 (17.9)
  Day 14: number analyzed (Participants) | 8 | 6
  Day 14 | 10540 (14.9) | 18400 (20.4)
Statistical Analysis 1: Comparison: Part 2: 30 mg S-648414 + Midazolam vs Part 2: 50 mg S-648414 + Midazolam; The dose proportionality of plasma S-648414 AUC0-τ after a single dose of S-648414 (Day 1) was assessed using an ANOVA model fitted to the ln-transformed AUC0-τ, with dose group fitted as a fixed factor. The point estimates and 90% CIs were generated for the ratios of the 50 mg dose to 30 mg dose ln-transformed AUC0-τ, then back-transformed to obtain the corresponding geometric least squares mean ratio and 90% CI; Test type: Other; Geometric Least Squares Mean Ratio = 1.6277, 90% CI 2-sided [1.4038 to 1.8874] — Ratio = 50 mg / 30 mg
Statistical Analysis 2: Comparison: Part 2: 30 mg S-648414 + Midazolam vs Part 2: 50 mg S-648414 + Midazolam; The dose proportionality of plasma S-648414 AUC0-τ after multiple doses of S-648414 (Day 14) was assessed using an ANOVA model fitted to the ln-transformed AUC0-τ, with dose group fitted as a fixed factor. The point estimates and 90% CIs were generated for the ratios of the 50 mg dose to 30 mg dose ln-transformed AUC0-τ, then back-transformed to obtain the corresponding geometric least squares mean ratio and 90% CI; Test type: Other; Geometric Least Squares Mean Ratio = 1.7454, 90% CI 2-sided [1.4785 to 2.0605] — Ratio = 50 mg / 30 mg
Statistical Analysis 3: Comparison: Part 2: 30 mg S-648414 + Midazolam; The accumulation ratio of AUC0-τ in the 30 mg dose group was calculated as the ratio of Day 14 to Day 1 using an ANOVA fitted with a linear mixed model with ln-transformed AUC0-τ, Day as a fixed effect and participant as a random effect. The difference and 90% CI between the ln-transformed AUC0-τ on Day 1 and Day 14 were estimated then back-transformed to obtain the corresponding geometric least squares mean ratio and 90% CI; Test type: Other; Geometric Least Squares Mean Ratio = 1.9102, 90% CI 2-sided [1.7788 to 2.0513] — Ratio = Day 14 / Day 1
Statistical Analysis 4: Comparison: Part 2: 50 mg S-648414 + Midazolam; The accumulation ratio of AUC0-τ in the 50 mg dose group was calculated as the ratio of Day 14 to Day 1 using an ANOVA fitted with a linear mixed model with ln-transformed AUC0-τ, Day as a fixed effect and participant as a random effect. The difference and 90% CI between the ln-transformed AUC0-τ on Day 1 and Day 14 were estimated then back-transformed to obtain the corresponding geometric least squares mean ratio and 90% CI; Test type: Other; Geometric Least Squares Mean Ratio = 2.0478, 90% CI 2-sided [1.9203 to 2.1837] — Ratio = Day 14 / Day 1

28. Secondary Outcome: Part 2: Terminal Elimination Half-life (t1/2,z) of S-648414 Following Multiple-dose Administration
Description: Terminal elimination half-life, where t1/2,z = (ln2)/λz on Day 14.
Time Frame: Day 14 predose (0 hours), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, and 96 hours postdose.
Population: The PK parameter population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 2: 30 mg S-648414 + Midazolam | Part 2: 50 mg S-648414 + Midazolam
Number analyzed (Participants) | 8 | 6
hours | 21.6 (12.5) | 23.7 (11.0)

29. Secondary Outcome: Part 2: Terminal Elimination Rate Constant (λz) of S-648414 Following Multiple-dose Administration
Description: Terminal elimination rate constant, where λz is the magnitude of the slope of the linear regression of the log concentration versus time profile during the terminal phase on Day 14.
Time Frame: Day 14 predose (0 hours), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, and 96 hours postdose.
Population: The PK parameter population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hours
Arm/Group | Part 2: 30 mg S-648414 + Midazolam | Part 2: 50 mg S-648414 + Midazolam
Number analyzed (Participants) | 8 | 6
1/hours | 0.0321 (12.5) | 0.0292 (11.0)

30. Secondary Outcome: Part 2: Apparent Total Clearance (CL/F) of S-648414 Following Multiple-dose Administration
Description: Apparent total clearance estimated according to: CL/F = Dose/AUC0-τ on Day 14
Time Frame: Day 14 predose (0 hours), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours postdose.
Population: The PK parameter population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Part 2: 30 mg S-648414 + Midazolam | Part 2: 50 mg S-648414 + Midazolam
Number analyzed (Participants) | 8 | 6
L/hr | 2.85 (14.9) | 2.72 (20.4)

31. Secondary Outcome: Part 2: Apparent Volume of Distribution in the Terminal Elimination Phase (Vz/F) of S-648414 Following Multiple-dose Administration
Description: Apparent volume of distribution in the terminal elimination phase on Day 14, estimated according to: Vz /F = Dose/AUC0-τ/λz
Time Frame: Day 14 predose (0 hours), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, and 96 hours postdose.
Population: The PK parameter population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Part 2: 30 mg S-648414 + Midazolam | Part 2: 50 mg S-648414 + Midazolam
Number analyzed (Participants) | 8 | 6
liters | 88.7 (13.6) | 93.0 (28.5)

32. Secondary Outcome: Part 2: Fraction of S-648414 Dose Excreted in Urine Over the Dosing Interval (Feu0- τ) Following Multiple-dose Administration
Description: Fraction of dose excreted in urine over the dosing interval τ (24 hours) on Day 14 calculated as Aeu0-τ/Dose × 100, where Aeu0-τ is the amount of drug excreted in urine over the dosing interval τ (24 hours).
Time Frame: Day 14 0-24 hours postdose
Population: The PK parameter population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent excreted
Arm/Group | Part 2: 30 mg S-648414 + Midazolam | Part 2: 50 mg S-648414 + Midazolam
Number analyzed (Participants) | 8 | 6
percent excreted | 33.3 (15.7) | 35.0 (25.6)

33. Secondary Outcome: Part 2: Renal Clearance (CLR) of S-648414 Following Multiple-dose Administration
Description: Renal clearance on Day 14, calculated as CLR = Aeu0-τ/AUC0-τ, where Aeu0-τ is the amount of drug excreted in urine over the dosing interval τ (24 hours)
Time Frame: Day 14 0-24 hours postdose
Population: The PK parameter population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Part 2: 30 mg S-648414 + Midazolam | Part 2: 50 mg S-648414 + Midazolam
Number analyzed (Participants) | 8 | 6
L/hr | 0.948 (18.4) | 0.952 (18.1)

34. Secondary Outcome: Part 2: Maximum Plasma Concentration (Cmax) of Midazolam
Description: The effect of S-648414 on the PK of midazolam (a cytochrome P450 3A [CYP3A] substrate) was assessed in Part 2 following 5 mg midazolam administration alone (Day -2) and co-administration with S-648414 30 or 50 mg (Day 14).
Time Frame: Day -2 and Day 14 predose (0 hours), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours postdose.
Population: The PK parameter population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part 2: Midazolam (30 mg S-648414 Group): Participants assigned to the 30 mg S-648414 dose group received a single oral dose of 5 mg midazolam on Day -2
- Part 2: 30 mg S-648414 + Midazolam: Participants received 30 mg S-648414 and a single oral dose of 5 mg midazolam on Day 14.
- Part 2: Midazolam (50 mg S-648414 Group): Participants assigned to the 50 mg S-648414 dose group received a single oral dose of 5 mg midazolam on Day -2
- Part 2: 50 mg S-648414 + Midazolam: Participants received 50 mg S-648414 and a single oral dose of 5 mg midazolam on Day 14.
Arm/Group | Part 2: Midazolam (30 mg S-648414 Group) | Part 2: 30 mg S-648414 + Midazolam | Part 2: Midazolam (50 mg S-648414 Group) | Part 2: 50 mg S-648414 + Midazolam
Number analyzed (Participants) | 8 | 8 | 8 | 6
ng/mL | 18.0 (33.6) | 16.8 (25.6) | 19.5 (30.6) | 19.3 (33.2)
Statistical Analysis 1: Comparison: Part 2: Midazolam (30 mg S-648414 Group) vs Part 2: 30 mg S-648414 + Midazolam; The effect of S-648414 on the PK of midazolam (a CYP3A substrate) was assessed using an ANOVA fitted with a linear mixed effect model with ln-transformed Cmax as the dependent variable, treatment as a fixed effect, and participant as a random effect. The difference and 90% CI between the ln-transformed Cmax of midazolam plus S-648414 and midazolam alone was estimated then back-transformed to obtain the corresponding geometric least squares mean ratios and 90% CIs; Test type: Other — The drug interaction was assessed by whether the 90% CIs for the geometric least squares mean ratio of Cmax, AUC0-last, and AUC0-inf of midazolam were completely contained within the range of 0.8000 to 1.2500; Geometric Least Squares Mean Ratio = 0.9241, 90% CI 2-sided [0.8057 to 1.0600] — Ratio = 30 mg S-648414 + Midazolam / Midazolam
Statistical Analysis 2: Comparison: Part 2: Midazolam (50 mg S-648414 Group) vs Part 2: 50 mg S-648414 + Midazolam; [analysis description as in outcome 34, analysis 1]; Test type: Other — [test comment as in outcome 34, analysis 1]; Geometric Least Squares Mean Ratio = 1.0303, 90% CI 2-sided [0.9299 to 1.1415] — Ratio = 50 mg S-648414 + Midazolam / Midazolam

35. Secondary Outcome: Part 2: Time to Maximum Plasma Concentration of Midazolam
Description: as for outcome 34
Time Frame: Day -2 and Day 14 predose (0 hours), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours postdose.
Population: The PK parameter population with available data
Measure: Median (Full Range); unit: hours
Arm/Group | Part 2: Midazolam (30 mg S-648414 Group) | Part 2: 30 mg S-648414 + Midazolam | Part 2: Midazolam (50 mg S-648414 Group) | Part 2: 50 mg S-648414 + Midazolam
Number analyzed (Participants) | 8 | 8 | 8 | 6
hours | 0.76 [0.50 to 2.00] | 1.00 [0.50 to 2.08] | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 1.00]

36. Secondary Outcome: Part 2: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration After Dosing (AUC0-last) for Midazolam
Description: The effect of S-648414 on the PK of midazolam (a cytochrome P450 3A [CYP3A] substrate) was assessed in Part 2 following 5 mg midazolam administration alone (Day -2) and co-administration with S-648414 30 or 50 mg (Day 14).
  Area under the concentration-time curve from time zero to the time of the last quantifiable concentration after dosing, calculated by linear up/log down trapezoidal method.
Time Frame: Day -2 and Day 14 predose (0 hours), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours postdose.
Population: The PK parameter population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 2: Midazolam (30 mg S-648414 Group) | Part 2: 30 mg S-648414 + Midazolam | Part 2: Midazolam (50 mg S-648414 Group) | Part 2: 50 mg S-648414 + Midazolam
Number analyzed (Participants) | 8 | 8 | 8 | 6
ng*hr/mL | 70.17 (30.7) | 59.83 (40.5) | 73.28 (40.7) | 64.53 (35.6)
Statistical Analysis 1: Comparison: Part 2: Midazolam (30 mg S-648414 Group) vs Part 2: 30 mg S-648414 + Midazolam; The effect of S-648414 on the PK of midazolam (a CYP3A substrate) was assessed using an ANOVA fitted with a linear mixed effect model with ln-transformed AUC0-last as the dependent variable, treatment as a fixed effect, and participant as a random effect. The difference and 90% CI between the ln-transformed AUC0-last of midazolam plus S-648414 and midazolam alone was estimated then back-transformed to obtain the corresponding geometric least squares mean ratios and 90% CIs; Test type: Other — [test comment as in outcome 34, analysis 1]; Geometric Least Squares Mean Ratio = 0.8420, 90% CI 2-sided [0.6628 to 1.0696] — Ratio = 30 mg S-648414 + Midazolam / Midazolam
Statistical Analysis 2: Comparison: Part 2: Midazolam (50 mg S-648414 Group) vs Part 2: 50 mg S-648414 + Midazolam; [analysis description as in outcome 36, analysis 1]; Test type: Other — [test comment as in outcome 34, analysis 1]; Geometric Least Squares Mean Ratio = 0.8542, 90% CI 2-sided [0.7185 to 1.0155] — Ratio = 50 mg S-648414 + Midazolam / Midazolam

37. Secondary Outcome: Part 2: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of Midazolam
Description: The effect of S-648414 on the PK of midazolam (a cytochrome P450 3A [CYP3A] substrate) was assessed in Part 2 following 5 mg midazolam administration alone (Day -2) and co-administration with S-648414 30 or 50 mg (Day 14).
  Area under the concentration-time curve extrapolated from time zero to infinity defined as AUC0-last + (Clast/λz), where Clast is the last measurable plasma concentration and λz is the plasma terminal elimination rate constant.
Time Frame: Day -2 and Day 14 predose (0 hours), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours postdose.
Population: The PK parameter population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 2: Midazolam (30 mg S-648414 Group) | Part 2: 30 mg S-648414 + Midazolam | Part 2: Midazolam (50 mg S-648414 Group) | Part 2: 50 mg S-648414 + Midazolam
Number analyzed (Participants) | 8 | 8 | 8 | 6
ng*hr/mL | 72.81 (28.7) | 61.68 (41.2) | 76.03 (42.2) | 67.02 (37.1)
Statistical Analysis 1: Comparison: Part 2: Midazolam (30 mg S-648414 Group) vs Part 2: 30 mg S-648414 + Midazolam; The effect of S-648414 on the PK of midazolam (a CYP3A substrate) was assessed using an ANOVA fitted with a linear mixed effect model with ln-transformed AUC0-inf as the dependent variable, treatment as a fixed effect, and participant as a random effect. The difference and 90% CI between the ln-transformed AUC0-inf of midazolam plus S-648414 and midazolam alone was estimated then back-transformed to obtain the corresponding geometric least squares mean ratios and 90% CIs; Test type: Other — [test comment as in outcome 34, analysis 1]; Geometric Least Squares Mean Ratio = 0.8377, 90% CI 2-sided [0.6645 to 1.0561] — Ratio = 30 mg S-648414 + Midazolam / Midazolam
Statistical Analysis 2: Comparison: Part 2: Midazolam (50 mg S-648414 Group) vs Part 2: 50 mg S-648414 + Midazolam; [analysis description as in outcome 37, analysis 1]; Test type: Other — [test comment as in outcome 34, analysis 1]; Geometric Least Squares Mean Ratio = 0.8529, 90% CI 2-sided [0.7213 to 1.0085] — Ratio = 50 mg S-648414 + Midazolam / Midazolam

38. Secondary Outcome: Part 2: Terminal Elimination Half-life for Midazolam
Description: as for outcome 34
Time Frame: Day -2 and Day 14 predose (0 hours), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours postdose.
Population: The PK parameter population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 2: Midazolam (30 mg S-648414 Group) | Part 2: 30 mg S-648414 + Midazolam | Part 2: Midazolam (50 mg S-648414 Group) | Part 2: 50 mg S-648414 + Midazolam
Number analyzed (Participants) | 8 | 8 | 8 | 6
hours | 5.07 (18.7) | 4.64 (32.4) | 4.41 (41.1) | 4.54 (39.5)

39. Secondary Outcome: Part 2: Terminal Elimination Rate Constant for Midazolam
Description: as for outcome 34
Time Frame: Day -2 and Day 14 predose (0 hours), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours postdose.
Population: The PK parameter population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Part 2: Midazolam (30 mg S-648414 Group) | Part 2: 30 mg S-648414 + Midazolam | Part 2: Midazolam (50 mg S-648414 Group) | Part 2: 50 mg S-648414 + Midazolam
Number analyzed (Participants) | 8 | 8 | 8 | 6
1/hour | 0.1366 (18.7) | 0.1494 (32.4) | 0.1570 (41.1) | 0.1528 (39.5)

40. Secondary Outcome: Part 2: Mean Residence Time for Midazolam
Description: The effect of S-648414 on the PK of midazolam (a cytochrome P450 3A [CYP3A] substrate) was assessed in Part 2 following 5 mg midazolam administration alone (Day -2) and co-administration with S-648414 30 or 50 mg (Day 14).
  Mean residence time was calculated as MRT = AUMC0-inf/AUC0-inf where AUMC0-inf is the area under the first moment curve extrapolated to infinity.
Time Frame: Day -2 and Day 14 predose (0 hours), 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, and 24 hours postdose.
Population: The PK parameter population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 2: Midazolam (30 mg S-648414 Group) | Part 2: 30 mg S-648414 + Midazolam | Part 2: Midazolam (50 mg S-648414 Group) | Part 2: 50 mg S-648414 + Midazolam
Number analyzed (Participants) | 8 | 8 | 8 | 6
hours | 5.30 (8.6) | 4.44 (28.3) | 4.93 (33.8) | 4.40 (38.0)

41. Secondary Outcome: Part 1: Change From Baseline in Fridericia's Corrected QT Interval (QTcF)
Description: Continuous 12-lead digital electrocardiogram (ECG) recording was performed on Day 1. The QT interval is a measure between Q and T wave in heart's electrical cycle. ECGs were analyzed at a blinded, central ECG laboratory. At each specified time point, ten 14-second 12-lead ECG tracings were extracted from the continuous recordings. The median QT in each replicate was calculated; the mean of available medians was used as the participant's reportable value at that time point.
  QT interval was corrected for heart rate using Fridericia's correction (QTcF). Baseline was defined as the average of the measured ECG intervals from the 3 pre-dose time points (45, 30, and 15 minutes before dosing) on Day 1.
  Change from Baseline (ΔQTcF) was calculated based on a linear mixed-effects model with time (categorical), treatment, and time-by-treatment interaction as fixed effects and Baseline QTcF as covariate.
Time Frame: Day 1: Predose at 3 time points (-45, -30 and -15 minutes), and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours postdose.
Population: The QT/QTc population included all study participants randomly assigned to study intervention and who took at least 1 dose of study intervention.who had measurements at Baseline as well as on-treatment, with at least 1 post-dose time point with a valid ΔQTcF value. Participants with available data at each time point are included. Cardiodynamic ECG assessments were performed for Part 1 only.
Measure: Least Squares Mean (Standard Error); unit: ms
Groups:
- Part 1: 100 mg S-648414: Participants received a single oral dose of 100 mg S-648414 in a fasted state on Day 1.
Arm/Group | Part 1: Placebo | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 12 | 6 | 6 | 8 | 6 | 6 | 6
ms
  0.5 hours postdose | -3.2 (1.16) | -3.2 (1.61) | -5.6 (1.61) | -4.8 (1.40) | -4.1 (1.64) | -5.6 (1.69) | 2.0 (1.62)
  1 hour postdose | -2.2 (1.19) | -0.4 (1.66) | -2.4 (1.66) | -3.2 (1.44) | -0.9 (1.69) | -1.0 (1.74) | 4.9 (1.67)
  1.5 hours postdose | -1.1 (1.40) | -1.2 (1.96) | -2.6 (1.96) | -1.1 (1.69) | 1.8 (1.98) | 3.1 (2.02) | 4.9 (1.96)
  2 hours postdose | -0.1 (1.38) | -2.1 (1.93) | -1.0 (1.93) | -1.9 (1.67) | -1.2 (1.95) | 2.4 (1.99) | 6.3 (1.93)
  2.5 hours postdose | -2.5 (1.39) | -1.7 (1.94) | -1.5 (1.94) | -1.1 (1.68) | 0.4 (1.97) | 2.5 (2.01) | 8.0 (1.95)
  3 hours postdose | -1.9 (1.24) | 2.3 (1.73) | -1.3 (1.73) | -0.6 (1.50) | 2.6 (1.76) | -0.4 (1.80) | 10.1 (1.74)
  4 hours postdose | -2.3 (1.54) | -0.2 (2.16) | -0.6 (2.16) | 0.1 (1.87) | 0.2 (2.18) | 3.6 (2.22) | 12.0 (2.17)
  6 hours postdose | -5.3 (2.52) | -12.0 (3.55) | -2.3 (3.56) | -1.2 (3.08) | -4.6 (3.57) | -4.6 (3.59) | 2.9 (3.56)
  8 hours postdose | -4.1 (1.71) | -6.7 (2.41) | -0.3 (2.41) | -3.2 (2.08) | -5.9 (2.43) | -3.4 (2.46) | 5.0 (2.41)
  12 hours postdose | -0.9 (2.44) | -1.8 (3.44) | 0.9 (3.44) | 1.0 (2.98) | -1.3 (3.45) | -3.0 (3.48) | 8.8 (3.44)
  24 hours postdose: number analyzed (Participants) | 12 | 6 | 6 | 8 | 6 | 6 | 4
  24 hours postdose | -1.4 (1.19) | -4.9 (1.66) | -1.2 (1.66) | -2.1 (1.44) | -0.8 (1.69) | -1.8 (1.74) | 7.5 (2.01)

42. Secondary Outcome: Parts 1: Change From Baseline in Heart Rate (HR)
Description: Continuous 12-lead digital electrocardiogram (ECG) recording was performed on Day 1. ECGs were analyzed at a blinded, central ECG laboratory. At each specified time point, ten 14-second 12-lead ECG tracings were extracted from the continuous recordings. The median HR in each replicate was calculated; the mean of available medians was used as the participant's reportable value at that time point.
  Baseline was defined as the average of the measured ECG values from the 3 pre-dose time points (45, 30, and 15 minutes before dosing) on Day 1.
  Change from Baseline in HR (ΔHR) was calculated based on a linear mixed-effects model with time (categorical), treatment, and time-by-treatment interaction as fixed effects and Baseline HR as covariate.
Time Frame: as for outcome 41
Population: The QT/QTc population with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Part 1: Placebo | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 12 | 6 | 6 | 8 | 6 | 6 | 6
beats per minute
  0.5 hours postdose | 0.9 (1.11) | -0.2 (1.58) | -1.4 (1.60) | -1.1 (1.36) | -0.1 (1.57) | -0.7 (1.57) | -1.6 (1.57)
  1 hour postdose | 1.5 (1.16) | -2.7 (1.64) | -1.9 (1.66) | -2.1 (1.41) | 0.4 (1.64) | -1.0 (1.63) | -0.8 (1.63)
  1.5 hours postdose | -0.4 (1.18) | -3.0 (1.67) | -0.3 (1.69) | -3.0 (1.44) | -0.5 (1.67) | 0.2 (1.67) | -0.4 (1.66)
  2 hours postdose | -0.5 (1.30) | -3.2 (1.85) | -2.4 (1.87) | -2.5 (1.60) | -1.7 (1.85) | 0.4 (1.85) | -0.3 (1.84)
  2.5 hours postdose | 0.8 (1.28) | -1.2 (1.82) | -3.0 (1.84) | -2.2 (1.57) | -0.7 (1.81) | 2.7 (1.81) | -0.7 (1.81)
  3 hours postdose | -0.9 (1.38) | -3.0 (1.96) | -1.6 (1.97) | -2.1 (1.69) | -1.8 (1.95) | 2.0 (1.95) | -0.6 (1.95)
  4 hours postdose | 0.2 (1.41) | -1.2 (2.00) | 0.7 (2.02) | -2.8 (1.73) | 0.8 (2.00) | 2.1 (2.00) | 3.3 (2.00)
  6 hours postdose | 5.2 (1.18) | 4.6 (1.68) | 2.4 (1.70) | 4.2 (1.45) | 3.7 (1.67) | 7.3 (1.67) | 7.5 (1.67)
  8 hours postdose | 1.5 (1.56) | 1.7 (2.21) | 0.7 (2.22) | -0.2 (1.91) | 1.8 (2.20) | 4.6 (2.20) | 3.5 (2.20)
  12 hours postdose | 2.7 (1.80) | 1.1 (2.55) | 1.9 (2.56) | 1.1 (2.21) | 2.4 (2.55) | 9.1 (2.55) | 3.4 (2.55)
  24 hours postdose: number analyzed (Participants) | 12 | 6 | 6 | 8 | 6 | 6 | 4
  24 hours postdose | 0.4 (1.64) | -1.7 (2.33) | -0.4 (2.34) | -1.4 (2.01) | 0.8 (2.33) | 0.3 (2.32) | 3.3 (2.59)

43. Secondary Outcome: Part 1: Change From Baseline in PR Interval
Description: Continuous 12-lead digital electrocardiogram (ECG) recording was performed on Day 1. The PR interval is the time from the onset of the P-wave to the start of the next QRS complex. ECGs were analyzed at a blinded, central ECG laboratory. At each specified time point, ten 14-second 12-lead ECG tracings were extracted from the continuous recordings. The median PR in each replicate was calculated; the mean of available medians was used as the participant's reportable value at that time point.
  Baseline was defined as the average of the measured ECG intervals from the 3 pre-dose time points (45, 30, and 15 minutes before dosing) on Day 1.
  Change from Baseline in PR interval (ΔPR) was calculated based on a linear mixed-effects model with time (categorical), treatment, and time-by-treatment interaction as fixed effects and Baseline PR as covariate.
Time Frame: as for outcome 41
Population: The QT/QTc population with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: ms
Arm/Group | Part 1: Placebo | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 12 | 6 | 6 | 8 | 6 | 6 | 6
ms
  0.5 hours postdose | 0.4 (1.29) | 1.0 (1.87) | 2.2 (1.83) | -0.1 (1.61) | 1.3 (1.85) | -3.9 (1.84) | 0.0 (1.83)
  1 hour postdose | 0.9 (1.29) | 1.0 (1.86) | 4.0 (1.82) | 1.3 (1.60) | 1.9 (1.84) | -6.4 (1.83) | 1.0 (1.82)
  1.5 hours postdose | 0.4 (1.74) | 3.4 (2.49) | 1.0 (2.46) | 0.9 (2.15) | 2.2 (2.47) | 0.8 (2.47) | 0.9 (2.46)
  2 hours postdose | 0.8 (1.44) | 2.8 (2.07) | 3.4 (2.03) | -2.3 (1.78) | -1.4 (2.05) | -2.1 (2.04) | 0.2 (2.04)
  2.5 hours postdose | 0.7 (1.60) | 1.1 (2.29) | 4.5 (2.26) | -0.1 (1.97) | 0.5 (2.27) | -5.2 (2.26) | -0.9 (2.26)
  3 hours postdose | -0.1 (1.86) | 3.6 (2.67) | 3.7 (2.64) | 1.7 (2.30) | -1.5 (2.65) | -5.3 (2.64) | -0.7 (2.64)
  4 hours postdose | 0.5 (1.67) | 3.0 (2.39) | 3.1 (2.36) | -1.0 (2.06) | -0.1 (2.37) | -6.9 (2.36) | -1.7 (2.36)
  6 hours postdose | -2.8 (1.56) | -1.6 (2.24) | 0.7 (2.21) | -2.3 (1.93) | -0.9 (2.22) | -7.0 (2.21) | -3.0 (2.21)
  8 hours postdose | -3.2 (1.90) | -1.8 (2.71) | 3.6 (2.68) | -4.5 (2.34) | -5.8 (2.69) | -5.8 (2.69) | -1.8 (2.68)
  12 hours postdose | -0.9 (2.12) | 0.4 (3.03) | 3.5 (3.00) | -1.3 (2.61) | -1.0 (3.01) | -7.8 (3.01) | -0.5 (3.01)
  24 hours postdose: number analyzed (Participants) | 12 | 6 | 6 | 8 | 6 | 6 | 4
  24 hours postdose | -1.5 (1.61) | 0.1 (2.32) | 0.8 (2.28) | 0.5 (1.99) | -4.2 (2.29) | -2.2 (2.29) | -3.1 (2.52)

44. Secondary Outcome: Part 1: Change From Baseline in QRS Interval
Description: Continuous 12-lead digital electrocardiogram (ECG) recording was performed on Day 1. The QRS complex is a combination of the Q wave, R wave and S wave on an ECG tracing, and represents ventricular depolarization. ECGs were analyzed at a blinded, central ECG laboratory. At each specified time point, ten 14-second 12-lead ECG tracings were extracted from the continuous recordings. The median QRS in each replicate was calculated; the mean of available medians was used as the participant's reportable value at that time point.
  Baseline was defined as the average of the measured ECG intervals from the 3 pre-dose time points (45, 30, and 15 minutes before dosing) on Day 1.
  Change from Baseline in QRS interval (ΔQRS) was calculated based on a linear mixed-effects model with time (categorical), treatment, and time-by-treatment interaction as fixed effects and Baseline QRS as covariate.
Time Frame: as for outcome 41
Population: The QT/QTc population with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: ms
Arm/Group | Part 1: Placebo | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 12 | 6 | 6 | 8 | 6 | 6 | 6
ms
  0.5 hours postdose | -0.3 (0.21) | 0.0 (0.31) | -0.4 (0.30) | 0.2 (0.26) | -0.1 (0.31) | 0.1 (0.30) | -.1 (0.31)
  1 hour postdose | -0.4 (0.22) | -0.1 (0.32) | 0.1 (0.32) | 0.2 (0.27) | 0.3 (0.32) | 0.2 (0.32) | 0.4 (0.32)
  1.5 hours postdose | 0.5 (0.45) | -0.2 (0.63) | 0.0 (0.63) | 0.4 (0.55) | 0.5 (0.63) | 0.3 (0.63) | 0.6 (0.63)
  2 hours postdose | -0.3 (0.24) | 0.2 (0.34) | 0.1 (0.34) | 0.7 (0.29) | 0.1 (0.34) | 0.4 (0.34) | 0.8 (0.34)
  2.5 hours postdose | -0.1 (0.24) | 0.0 (0.34) | 0.2 (0.34) | -0.2 (0.30) | 0.2 (0.34) | 0.0 (0.34) | 0.3 (0.34)
  3 hours postdose | -0.2 (0.22) | 0.0 (0.31) | 0.2 (0.31) | 0.1 (0.27) | 0.4 (0.31) | 0.4 (0.31) | 0.2 (0.31)
  4 hours postdose | 0.2 (0.29) | -0.1 (0.41) | 0.2 (0.41) | 0.5 (0.35) | 0.3 (0.41) | 0.9 (0.41) | 1.0 (0.41)
  6 hours postdose | -0.5 (0.55) | -0.8 (0.78) | -0.5 (0.77) | -0.7 (0.67) | -1.3 (0.78) | 0.6 (0.77) | 0.8 (0.78)
  8 hours postdose | -0.8 (0.33) | -0.6 (0.47) | -0.2 (0.47) | -0.3 (0.41) | -0.3 (0.47) | 0.2 (0.47) | -0.5 (0.47)
  12 hours postdose | -1.4 (0.38) | 0.0 (0.54) | 0.0 (0.54) | -0.3 (0.47) | -0.3 (0.54) | 0.5 (0.54) | 0.5 (0.54)
  24 hours postdose: number analyzed (Participants) | 12 | 6 | 6 | 8 | 6 | 6 | 4
  24 hours postdose | -0.7 (0.39) | 0.1 (0.55) | 0.1 (0.55) | 0.4 (0.48) | -0.1 (0.55) | 0.0 (0.55) | -0.7 (0.64)

45. Secondary Outcome: Part 1: Placebo-corrected Change From Baseline in Fridericia's Corrected QT Interval
Description: Continuous 12-lead digital electrocardiogram (ECG) recording was performed on Day 1. ECGs were analyzed at a blinded, central ECG laboratory. At each specified time point, ten 14-second 12-lead ECG tracings were extracted from the continuous recordings. The median QT in each replicate was calculated; the mean of available medians was used as the participant's reportable value at that time point.
  QT interval was corrected for heart rate using Fridericia's correction (QTcF). Baseline was defined as the average of the measured ECG intervals from the 3 pre-dose time points (45, 30, and 15 minutes before dosing) on Day 1.
  Change from Baseline (ΔQTcF) was calculated based on a linear mixed-effects model with time (categorical), treatment, and time-by-treatment interaction as fixed effects and Baseline QTcF as covariate.
  Placebo-corrected ΔQTcF (ΔΔQTcF) was calculated as the adjusted mean ΔQTcF in the S-648414 group minus adjusted mean ΔQTcF in the placebo group at each time point.
Time Frame: as for outcome 41
Population: The QT/QTc population with available data at each time point. The number of participants analyzed includes participants in each S-648414 group with available data; reported values are corrected for placebo data collected for the 12 participants in the Part 1 Placebo group.
Measure: Least Squares Mean (Standard Error); unit: ms
Arm/Group | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 6 | 6
ms
  0.5 hours postdose | 0.0 (1.98) | -2.4 (1.99) | -1.6 (1.81) | -0.9 (1.98) | -2.4 (2.10) | 5.2 (2.00)
  1 hour postdose | 1.7 (2.04) | -0.2 (2.06) | -1.0 (1.87) | 1.2 (2.04) | 1.1 (2.16) | 7.0 (2.07)
  1.5 hours postdose | -0.1 (2.40) | -1.5 (2.41) | 0.0 (2.20) | 3.0 (2.40) | 4.2 (2.50) | 6.0 (2.42)
  2 hours postdose | -2.0 (2.37) | -0.9 (2.38) | -1.8 (2.16) | -1.1 (2.36) | 2.5 (2.46) | 6.4 (2.39)
  2.5 hours postdose | 0.8 (2.38) | 1.0 (2.39) | 1.4 (2.18) | 2.8 (2.38) | 5.0 (2.48) | 10.4 (2.40)
  3 hours postdose | 4.1 (2.13) | 0.5 (2.14) | 1.2 (1.94) | 4.5 (2.12) | 1.4 (2.24) | 12.0 (2.15)
  4 hours postdose | 2.1 (2.65) | 1.7 (2.66) | 2.4 (2.42) | 2.5 (2.65) | 5.9 (2.74) | 14.3 (2.67)
  6 hours postdose | -6.7 (4.36) | 3.0 (4.36) | 4.0 (3.98) | 0.7 (4.36) | 0.6 (4.41) | 8.1 (4.37)
  8 hours postdose | -2.7 (2.95) | 3.7 (2.96) | 0.9 (2.70) | -1.8 (2.95) | 0.7 (3.03) | 9.1 (2.97)
  12 hours postdose | -1.0 (4.21) | 1.8 (4.22) | 1.8 (3.85) | -0.5 (4.21) | -2.1 (4.27) | 9.6 (4.23)
  24 hours postdose: number analyzed (Participants) | 8 | 8 | 8 | 6 | 6 | 4
  24 hours postdose | -3.6 (2.04) | 0.2 (2.05) | -0.7 (1.86) | 0.5 (2.03) | -0.4 (2.15) | 8.8 (2.36)

46. Secondary Outcome: Part 1: Placebo-corrected Change From Baseline in Heart Rate
Description: Continuous 12-lead digital electrocardiogram (ECG) recording was performed on Day 1. ECGs were analyzed at a blinded, central ECG laboratory. At each specified time point, ten 14-second 12-lead ECG tracings were extracted from the continuous recordings. The median HR in each replicate was calculated; the mean of available medians was used as the participant's reportable value at that time point.
  Baseline was defined as the average of the measured values from the 3 pre-dose time points (45, 30, and 15 minutes before dosing) on Day 1.
  Change from Baseline (ΔHR) was calculated based on a linear mixed-effects model with time (categorical), treatment, and time-by-treatment interaction as fixed effects and Baseline HR as covariate.
  Placebo-corrected ΔHR (ΔΔHR) was calculated as the adjusted mean ΔHR in the S-648414 group minus adjusted mean ΔHR in the placebo group at each time point.
Time Frame: as for outcome 41
Population: as for outcome 45
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 6 | 6 | 8 | 6 | 6 | 6
beats per minute
  0.5 hours postdose | -1.1 (1.93) | -2.3 (1.95) | -2.0 (1.76) | -1.0 (1.92) | -1.6 (1.93) | -2.5 (1.92)
  1 hour postdose | -4.2 (2.00) | -3.4 (2.03) | -3.5 (1.83) | -1.1 (2.00) | -2.5 (2.00) | -2.2 (2.00)
  1.5 hours postdose | -2.6 (2.04) | 0.1 (2.07) | -2.6 (1.86) | 0.0 (2.04) | 0.6 (2.04) | 0.0 (2.04)
  2 hours postdose | -2.7 (2.26) | -2.0 (2.28) | -2.1 (2.06) | -1.3 (2.26) | 0.9 (2.26) | 0.1 (2.26)
  2.5 hours postdose | -2.0 (2.22) | -3.8 (2.25) | -3.0 (2.03) | -1.5 (2.22) | 2.0 (2.22) | -1.5 (2.22)
  3 hours postdose | -2.1 (2.39) | -0.7 (2.41) | -1.2 (2.18) | -0.8 (2.39) | 2.9 (2.39) | 0.4 (2.39)
  4 hours postdose | -1.4 (2.45) | 0.4 (2.47) | -3.1 (2.23) | 0.6 (2.45) | 1.9 (2.45) | 3.1 (2.45)
  6 hours postdose | -0.6 (2.05) | -2.8 (2.07) | -1.0 (1.87) | -1.5 (2.05) | 2.0 (2.05) | 2.3 (2.05)
  8 hours postdose | 0.1 (2.70) | -0.9 (2.72) | -1.7 (2.46) | 0.3 (2.70) | 3.1 (2.70) | 2.0 (2.70)
  12 hours postdose | -1.6 (3.12) | -0.7 (3.14) | -1.5 (2.85) | -0.3 (3.12) | 6.4 (3.12) | 0.7 (3.12)
  24 hours postdose: number analyzed (Participants) | 6 | 6 | 8 | 6 | 6 | 4
  24 hours postdose | -2.2 (2.85) | -0.9 (2.87) | -1.9 (2.60) | 0.4 (2.85) | -0.1 (2.85) | 2.9 (3.06)

47. Secondary Outcome: Part 1: Placebo-corrected Change From Baseline in PR Interval
Description: Continuous 12-lead digital electrocardiogram (ECG) recording was performed on Day 1. ECGs were analyzed at a blinded, central ECG laboratory. At each specified time point, ten 14-second 12-lead ECG tracings were extracted from the continuous recordings. The median PR interval in each replicate was calculated; the mean of available medians was used as the participant's reportable value at that time point.
  Baseline was defined as the average of the measured ECG intervals from the 3 pre-dose time points (45, 30, and 15 minutes before dosing) on Day 1.
  Change from Baseline (ΔPR) was calculated based on a linear mixed-effects model with time (categorical), treatment, and time-by-treatment interaction as fixed effects and Baseline PR as covariate.
  Placebo-corrected ΔPR (ΔΔPR) was calculated as the adjusted mean ΔPR in the S-648414 group minus adjusted mean ΔPR in the placebo group at each time point.
Time Frame: as for outcome 41
Population: as for outcome 45
Measure: Least Squares Mean (Standard Error); unit: ms
Arm/Group | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 6 | 6 | 8 | 6 | 6 | 6
ms
  0.5 hours postdose | 0.6 (2.28) | 1.8 (2.24) | -0.5 (2.06) | 0.9 (2.25) | -4.3 (2.25) | -0.4 (2.24)
  1 hour postdose | 0.2 (2.27) | 3.2 (2.23) | 0.5 (2.05) | 1.0 (2.24) | -7.2 (2.23) | 0.2 (2.23)
  1.5 hours postdose | 3.0 (3.04) | 0.6 (3.02) | 0.5 (2.76) | 1.8 (3.02) | 0.4 (3.02) | 0.5 (3.02)
  2 hours postdose | 2.0 (2.52) | 2.6 (2.49) | -3.1 (2.29) | -2.2 (2.50) | -2.9 (2.49) | -0.6 (2.49)
  2.5 hours postdose | 0.4 (2.79) | 3.8 (2.77) | -0.8 (2.54) | -0.2 (2.78) | -5.9 (2.77) | -1.6 (2.77)
  3 hours postdose | 3.8 (3.25) | 3.8 (3.23) | 1.8 (2.96) | -1.4 (3.24) | -5.2 (3.23) | -0.5 (3.23)
  4 hours postdose | 2.5 (2.91) | 2.7 (2.89) | -1.5 (2.65) | -0.5 (2.90) | -7.4 (2.89) | -2.2 (2.89)
  6 hours postdose | 1.2 (2.74) | 3.5 (2.71) | 0.5 (2.48) | 1.9 (2.72) | -4.1 (2.71) | -0.1 (2.71)
  8 hours postdose | 1.4 (3.31) | 6.8 (3.28) | -1.3 (3.01) | -2.6 (3.29) | -2.6 (3.29) | 1.4 (3.29)
  12 hours postdose | 1.3 (3.70) | 4.5 (3.68) | -0.4 (3.37) | -0.1 (3.69) | -6.9 (3.68) | 0.4 (3.68)
  24 hours postdose: number analyzed (Participants) | 6 | 6 | 8 | 6 | 6 | 4
  24 hours postdose | 1.6 (2.82) | 2.2 (2.79) | 2.0 (2.56) | -2.7 (2.80) | -0.7 (2.80) | -1.6 (2.99)

48. Secondary Outcome: Part 1: Placebo-corrected Change From Baseline in QRS Duration
Description: Continuous 12-lead digital electrocardiogram (ECG) recording was performed on Day 1. ECGs were analyzed at a blinded, central ECG laboratory. At each specified time point, ten 14-second 12-lead ECG tracings were extracted from the continuous recordings. The median QRS duration in each replicate was calculated; the mean of available medians was used as the participant's reportable value at that time point.
  Baseline was defined as the average of the measured ECG intervals from the 3 pre-dose time points (45, 30, and 15 minutes before dosing) on Day 1.
  Change from Baseline in QRS duration (ΔQRS) was calculated based on a linear mixed-effects model with time (categorical), treatment, and time-by-treatment interaction as fixed effects and Baseline QRS as covariate.
  Placebo-corrected ΔQRS (ΔΔQRS) was calculated as the adjusted mean ΔQRS in the S-648414 group minus adjusted mean ΔQRS in the placebo group at each time point.
Time Frame: as for outcome 41
Population: as for outcome 45
Measure: Least Squares Mean (Standard Error); unit: ms
Arm/Group | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 6 | 6 | 8 | 6 | 6 | 6
ms
  0.5 hours postdose | 0.2 (0.37) | -0.1 (0.37) | 0.5 (0.34) | 0.2 (0.37) | 0.4 (0.37) | 0.2 (0.37)
  1 hour postdose | 0.3 (0.39) | 0.5 (0.39) | 0.6 (0.35) | 0.7 (0.39) | 0.6 (0.39) | 0.8 (0.39)
  1.5 hours postdose | -0.7 (0.77) | -0.6 (0.77) | -0.1 (0.71) | -0.1 (0.77) | -0.3 (0.77) | 0.0 (0.77)
  2 hours postdose | 0.5 (0.42) | 0.4 (0.42) | 1.1 (0.38) | 0.5 (0.42) | 0.7 (0.42) | 1.1 (0.42)
  2.5 hours postdose | 0.1 (0.42) | 0.3 (0.42) | -0.1 (0.38) | 0.3 (0.42) | 0.1 (0.42) | 0.4 (0.42)
  3 hours postdose | 0.2 (0.38) | 0.4 (0.38) | 0.3 (0.35) | 0.5 (0.38) | 0.5 (0.38) | 0.3 (0.38)
  4 hours postdose | -0.3 (0.50) | 0.0 (0.50) | 0.3 (0.46) | 0.1 (0.50) | 0.8 (0.50) | 0.8 (0.50)
  6 hours postdose | -0.3 (0.95) | 0.0 (0.95) | -0.2 (0.87) | -0.8 (0.95) | 1.1 (0.95) | 1.3 (0.95)
  8 hours postdose | 0.2 (0.58) | 0.7 (0.58) | 0.5 (0.53) | 0.5 (0.58) | 1.1 (0.58) | 0.3 (0.58)
  12 hours postdose | 1.4 (0.66) | 1.4 (0.66) | 1.1 (0.60) | 1.1 (0.66) | 1.9 (0.66) | 1.9 (0.66)
  24 hours postdose: number analyzed (Participants) | 6 | 6 | 8 | 6 | 6 | 4
  24 hours postdose | 0.8 (0.68) | 0.8 (0.67) | 1.1 (0.62) | 0.6 (0.68) | 0.7 (0.67) | 0.0 (0.75)

49. Secondary Outcome: Part 1: Number of Participants With Recorded Outlier Values for QTcF, HR, PR, and QRS
Description: A participant was determined as an outlier if the following criteria (assessed separately) were met for the ECG intervals at any time point:
  QTcF:
  * Treatment-emergent value of > 450 and ≤ 480 ms when not present at Baseline (new onset)
  * Treatment-emergent value of > 480 and ≤ 500 ms when not present at Baseline (new onset)
  * Treatment-emergent value of > 500 ms when not present at Baseline (new onset)
  * Increase of QTcF (ΔQTcF) from Baseline of > 30 and ≤ 60 ms
  * Increase of QTcF from Baseline > 60 ms
  HR:
  * Decrease of HR from Baseline > 25% resulting in HR < 50 bpm
  * Increase of HR from Baseline > 25% resulting in HR > 100 bpm
  PR:
  * Increase of PR from Baseline > 25% resulting in PR > 200 ms
  QRS:
  * Increase of QRS from Baseline > 25% resulting in QRS > 120 ms
Time Frame: as for outcome 41
Population: QT/QTc population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 12 | 6 | 6 | 8 | 6 | 6 | 6
Participants
  QTcF > 450 and ≤ 480 ms | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF > 480 and ≤ 500 ms | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF > 500 ms | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ΔQTcF > 30 and ≤ 60 ms | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ΔQTcF > 60 ms | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HR < 50 (bpm) with a decrease in ΔHR > 25% | 0 | 1 | 0 | 0 | 0 | 0 | 0
  HR > 100 (bpm) with an increase in ΔHR > 25% | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR > 200 (ms) with an increase in ΔPR > 25% | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS > 120 (ms) with an increase in ΔQRS > 25% | 0 | 0 | 0 | 0 | 0 | 0 | 0

50. Secondary Outcome: Part 1: Number of Participants With Treatment-emergent Changes for T-wave Morphology and U-wave Presence
Description: T-wave abnormalities were categorized as follows:
  * Normal T wave: Any positive T wave not meeting any criterion below
  * Flat T wave: T amplitude < 1 mm (either positive or negative) including flat isoelectric line
  * Notched T wave (+): Presence of notch(es) of at least 0.05 mV amplitude on ascending or descending arm of the positive T wave
  * Biphasic: T wave that contains a second component with an opposite phase that is at least 0.1 mV deep (both positive/negative and negative/positive and polyphasic T waves included)
  * Normal T wave (-): T amplitude that is negative, without biphasic T wave or notches
  * Notched T wave (-): Presence of notch(es) of at least 0.05 mV amplitude on descending or ascending arm of the negative T wave
  * U waves: Presence of abnormal U waves
Time Frame: as for outcome 41
Population: QT/QTc population)
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414
Number analyzed (Participants) | 12 | 6 | 6 | 8 | 6 | 6 | 6
Participants
  Flat | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Notched (+) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Biphasic | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Normal (-) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Notched (-) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  U-Wave presence | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Part 1: From dosing on Day 1 or Day 14 up to 10 days post dose; Part 2: From the first dose up to 10 days after end of dosing (25 days); Part 3: From the first dose up to Day 36. A TEAE was summarized to a given treatment if the event onset/worsening occurred any time after the dose of that treatment and before the dose of the next treatment.
Groups:
- Part 1: Placebo - Fasted: Participants received a single oral dose of matching placebo in a fasted state on Day 1.
- Part 1: Placebo - Fed: Participants received a single dose of matching placebo in a fed state (after a high-fat meal) on Day 14.
- Part 1: 100 mg S-648414 Fed: Participants received a single oral dose of 100 mg S-648414 in a fed state (after a high-fat meal) on Day 14.
- Part 2: Placebo (Days 1-13): Participants received matching placebo to S-648414 once a day on Days 1 to 13.
- Part 2: 50 mg S-648414 (Days 1-13): Participants received 50 mg S-648414 once a day on Days 1 to 13.
- Part 2: 30 mg S-648414 (Days 1-13): Participants received 30 mg S-648414 once a day on Days 1 to 13.
- Part 3: Group I Dolutegravir: Participants received 50 mg dolutegravir orally once a day on Days 1 to 7.
- Part 3: Dolutegravir: Participants received 50 mg dolutegravir once a day on Days 1 to 7.
Arm/Group | Part 1: Placebo - Fasted | Part 1: Placebo - Fed | Part 1: 10 mg S-648414 | Part 1: 30 mg S-648414 | Part 1: 100 mg S-648414 Fasted | Part 1: 100 mg S-648414 Fed | Part 1: 250 mg S-648414 | Part 1: 500 mg S-648414 | Part 1: 1000 mg S-648414 | Part 2: Midazolam (Day -2) | Part 2: Placebo (Days 1-13) | Part 2: 50 mg S-648414 (Days 1-13) | Part 2: 30 mg S-648414 (Days 1-13) | Part 2: Placebo + Midazolam (Day 14) | Part 2: 50 mg S-648414 + Midazolam (Day 14) | Part 2: 30 mg S-648414 + Midazolam (Day 14) | Part 3: Group I Dolutegravir | Part 3: 100 mg S-648414 | Part 3: 100 mg S-648414 + Dolutegravir | Part 3: Dolutegravir | Part 3: 200 mg S-648414 | Part 3: 200 mg S-648414 + Dolutegravir
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/2 | 0/6 | 0/6 | 0/8 | 0/8 | 0/6 | 0/6 | 0/6 | 0/20 | 0/4 | 0/8 | 0/8 | 0/2 | 0/7 | 0/8 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/2 | 0/6 | 0/6 | 0/8 | 0/8 | 0/6 | 0/6 | 0/6 | 0/20 | 0/4 | 0/8 | 0/8 | 0/2 | 0/7 | 0/8 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 2/12 | 0/2 | 0/6 | 1/6 | 2/8 | 2/8 | 1/6 | 1/6 | 2/6 | 0/20 | 2/4 | 2/8 | 3/8 | 0/2 | 1/7 | 1/8 | 3/14 | 3/14 | 4/14 | 2/14 | 5/14 | 2/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo - Fasted (N=12) | Part 1: Placebo - Fed (N=2) | Part 1: 10 mg S-648414 (N=6) | Part 1: 30 mg S-648414 (N=6) | Part 1: 100 mg S-648414 Fasted (N=8) | Part 1: 100 mg S-648414 Fed (N=8) | Part 1: 250 mg S-648414 (N=6) | Part 1: 500 mg S-648414 (N=6) | Part 1: 1000 mg S-648414 (N=6) | Part 2: Midazolam (Day -2) (N=20) | Part 2: Placebo (Days 1-13) (N=4) | Part 2: 50 mg S-648414 (Days 1-13) (N=8) | Part 2: 30 mg S-648414 (Days 1-13) (N=8) | Part 2: Placebo + Midazolam (Day 14) (N=2) | Part 2: 50 mg S-648414 + Midazolam (Day 14) (N=7) | Part 2: 30 mg S-648414 + Midazolam (Day 14) (N=8) | Part 3: Group I Dolutegravir (N=14) | Part 3: 100 mg S-648414 (N=14) | Part 3: 100 mg S-648414 + Dolutegravir (N=14) | Part 3: Dolutegravir (N=14) | Part 3: 200 mg S-648414 (N=14) | Part 3: 200 mg S-648414 + Dolutegravir (N=14)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 1 | 1
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intraocular pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT04147715/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT04147715/SAP_001.pdf